CLINICAL TRIAL: NCT03975790
Title: Comparative Analysis of Outcomes Among Patients Initiating Xeljanz in Combination With Oral MTX Who Withdraw MTX Versus Continue MTX Using a United States Healthcare Claims Database
Brief Title: Comparative Analysis of Outcomes Among Patients Initiating Xeljanz in Combination With Oral MTX Who Withdraw MTX Versus Continue MTX
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921336
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Results first posted 2019-10-22 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Truven Health MarketScan Research Database: Compare treatment patterns including dosing, concomitant medication use, adherence, persistence, and switching among tofacitinb+MTX patients who withdraw MTX vs. persist with MTX or experience interrupted MTX

SUMMARY:
To address the objectives, a retrospective cohort design will be employed to evaluate patient characteristics, treatment patterns, medication effectiveness, and health care cost and utilization in RA patients newly initiating tofacitinib in combination with oral methotrexate (MTX)

ELIGIBILITY:
Inclusion Criteria:

* At least one claim for tofacitinib between 01 January 2014 and 31 January 2017 (the identification period).
* Presence of The International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9 CM) code for RA (in any position) during the one-year pre-index period or on the index date. ICD-9 = 714.0x-714.4x & 714.81 or ICD10 = M05.* & M06.0*-M06.3* or M06.8*-M06.9*.
* At least 18 years old as of the index date.

Exclusion Criteria:

* Patients with claims for other conditions for which biologics are used during the one-year pre-index period or on the index date: ankylosing spondylitis, Crohn's disease, psoriasis, psoriatic arthritis, or ulcerative colitis will be excluded from the study.
* Patients with evidence of the index medication during the one-year pre-index period will be removed from the analysis. Patients will be allowed to have been treated with other biologics approved for RA (Tumor-Necrosis Factor-alpha inhibitors (TNFi) [adalimumab (Humira), etanercept (Enbrel), certolizumab pegol (Cimzia), golimumab (Simponi), infliximab (Remicade)] and non-TNFi's with alternative mechanisms of action [abatacept (Orencia), and rituximab (Rituxan), anakinra (Kineret), tocilizumab (Actemra)]) during the one-year pre-index period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are privately insured and with Medicare Supplemental insurance
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921336

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was a retrospective population-based register study. Detailed data on each participant was retrieved from the Truven Health MarketScan Research Database and assessed in this study.
Groups:
- Methotrexate (MTX) + Tofacitinib: MTX Persistent: Rheumatoid arthritis (RA) diagnosed participants who were privately insured or under Medicare Supplemental insurance (from their employer), initiated tofacitinib in combination with MTX, orally, between 01 January 2014 to 31 January 2017 (identification period) with no gap of more than (>)60 days in MTX therapy (persistent) within 12 months post-index date, were included in the study and their information as per Truven Health MarketScan Research Database (from January 1, 2012 to January 2018) was assessed in this study. Index date defined as the date of first claim for tofacitinib by participants to their insurance provider during identification period.
- Methotrexate (MTX) + Tofacitinib: MTX Discontinued: RA diagnosed participants who were privately insured or under Medicare Supplemental insurance (from their employer), initiated tofacitinib in combination with MTX, orally, between 01 January 2014 to 31 January 2017 (identification period) with a gap of >60 days in MTX therapy (discontinued) within 12 months post-index date, were included in the study and their information as per Truven Health MarketScan Research Database (from January 1, 2012 to January 2018) was assessed in this study. Index date defined as the date of first claim for tofacitinib by participants to their insurance provider during identification period.
- Methotrexate (MTX) + Tofacitinib: MTX Interrupted: RA diagnosed participants who were privately insured or under Medicare Supplemental insurance (from their employer), initiated tofacitinib in combination with MTX, orally, between 01 January 2014 to 31 January 2017 (identification period) with a gap of >60 days with 1 or more subsequent prescription re-fills in MTX therapy (interrupted) within 12 months post-index date, were included in the study and their information as per Truven Health MarketScan Research Database (from January 1, 2012 to January 2018) was assessed in this study. Index date defined as the date of first claim for tofacitinib by participants to their insurance provider during identification period.
Period: Overall Study
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Started | 337 | 94 | 48
Completed | 337 | 94 | 48
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants included in the study.
Groups:
- Methotrexate (MTX) + Tofacitinib: MTX Persistent: RA diagnosed participants who were privately insured or under Medicare Supplemental insurance (from their employer), initiated tofacitinib in combination with MTX, orally, between 01 January 2014 to 31 January 2017 (identification period) with no gap of >60 days in MTX therapy (persistent) within 12 months post-index date, were included in the study and their information as per Truven Health MarketScan Research Database (from January 1, 2012 to January 2018) was assessed in this study. Index date defined as the date of first claim for tofacitinib by participants to their insurance provider during identification period.
- Total: Total of all reporting groups
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted | Total
Number analyzed (Participants) | 337 | 94 | 48 | 479
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.10 (10.37) | 55.02 (9.81) | 58.08 (9.43) | 56.09 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 82 | 35 | 386
  Male | 68 | 12 | 13 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants as Per Type of Insurance Plan
Description: Number of participants covered by type of insurance is reported. There were two types of insurance: 1) a private insurance plan, that is, one purchased by the participants, commercially available; 2) employer-provided insurance plan, that is, the participant's employer provided the insurance.
Time Frame: During pre-index period (12 months duration before the index date [Index date: date of first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years])
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  Private insurance plan | 36 | 13 | 9
  Insurance plan from employer | 301 | 81 | 39

2. Primary Outcome: Number of Participants in Each Geographic Region
Description: Number of participants enrolled in the study per geographic region of the United States (northeast; north central; south; west; unknown) is reported.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  Northeast Region | 81 | 25 | 10
  North Central Region | 76 | 17 | 14
  South Region | 150 | 47 | 21
  West Region | 29 | 5 | 3
  Unknown Region | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Biologic Disease Modifying Antirheumatic Drug (bDMARD) Use During Pre-Index Period
Description: Number of Participants with use of at least one bDMARD during pre-index period is reported. The bDMARD could have been any tumor-necrosis factor-alpha inhibitors (TNFi), any non-TNFi, adalimumab, certolizumab pegol, etanercept, golimumab, infliximab, anakinra, abatacept, tocilizumab or rituximab.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 225 | 59 | 31
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.4695, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7644, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.8316, Chi-squared

4. Primary Outcome: Number of Participants With Biologic Disease Modifying Antirheumatic Drug (bDMARD) Use During Variable Length Pre-Index Period
Description: Number of Participants with use of at least one bDMARD during variable length pre-index period is reported. The bDMARD could have been any TNFi, any non-TNFi, adalimumab, certolizumab pegol, etanercept, golimumab, infliximab, anakinra, abatacept, tocilizumab or rituximab. Variable-length pre-index period defined as the period from the participant's first date of enrollment in the database to the day before the index date. The date of enrollment had to be at least 1 year prior to the index date and depending on the participant, could have been as much as maximum of 5.2 years. The index date was the date of the first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During variable length pre-index period (1 year before the index date up to 5.2 years)
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 247 | 69 | 36
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.9829, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.8021, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.8376, Chi-squared

5. Primary Outcome: Mean Number of Biologic Disease Modifying Antirheumatic Drug (bDMARD) Received During Pre-Index Period
Description: Mean number of bDMARD received during pre-index period is reported. The bDMARD could have been any TNFi, any non-TNFi, adalimumab, certolizumab pegol, etanercept, golimumab, infliximab, anakinra, abatacept, tocilizumab or rituximab.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: bDMARD
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 225 | 59 | 31
bDMARD | 1.38 (0.59) | 1.31 (0.46) | 1.23 (0.50)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.2864, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1583, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4546, t-test

6. Primary Outcome: Mean Number of Biologic Disease Modifying Antirheumatic Drug (bDMARD) Received During Variable Length Pre-Index Period
Description: Mean number of bDMARD received during variable length pre-index period is reported. The bDMARD could have been any TNFi, any non-TNFi, adalimumab, certolizumab pegol, etanercept, golimumab, infliximab, anakinra, abatacept, tocilizumab or rituximab. Variable-length pre-index period defined as the period from the participant's first date of enrollment in the database to the day before the index date. The date of enrollment had to be at least 1 year prior to the index date and depending on the participant could have been as much as maximum of 5.2 years. The index date was the date of the first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During variable length pre-index period (1 year before the index date up to 5.2 years)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: bDMARD
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 247 | 69 | 36
bDMARD | 1.81 (0.87) | 1.55 (0.76) | 1.50 (0.61)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.0280, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0106, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7293, t-test

7. Primary Outcome: Number of Participants With Non-biologic Disease Modifying Antirheumatic Drug (NB-DMARD) Use During Pre-Index Period
Description: Number of Participants with NB-DMARD use during pre-index period is reported. The NB-DMARD could have been hydroxychloroquine, MTX oral, leflunomide, sulfasalazine, chloroquine, cyclosporine, thalidomide, azathioprine, cyclophosphamide, auranofin, aurothioglucose, gold sodium thiomalate, penicillamine, tacrolimus or minocycline.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 333 | 93 | 47
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.9215, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6078, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6258, Chi-squared

8. Primary Outcome: Number of Participants With Non-Biologic Disease Modifying Antirheumatic Drug (NB-DMARD) Use During Variable Length Pre-Index Period
Description: Number of Participants with NB-MARD use during variable length pre-index period is reported. The NB-DMARD could have been hydroxychloroquine, MTX oral, leflunomide, sulfasalazine, chloroquine, cyclosporine, thalidomide, azathioprine, cyclophosphamide, auranofin, aurothioglucose, gold sodium thiomalate, penicillamine, tacrolimus or minocycline. Variable-length pre-index period defined as the period from the participant's first date of enrollment in the database to the day before the index date. The date of enrollment had to be at least 1 year prior to the index date and depending on the participant could have been as much as maximum of 5.2 years. The index date was the date of the first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During variable length pre-index period (1 year before the index date up to 5.2 years)
Population: Analysis was performed on all participants included in the study. p-value could not be calculated for reporting groups with 100% response.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 334 | 94 | 48
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.3586, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.5117, Chi-squared

9. Primary Outcome: Mean Number of Non-Biologic Disease Modifying Antirheumatic Drug (NB-DMARD) Received During Pre-Index Period
Description: Mean number of NB-DMARD received during pre-index period is reported. The NB-DMARD could have been hydroxychloroquine, MTX oral, leflunomide, sulfasalazine, chloroquine, cyclosporine, thalidomide, azathioprine, cyclophosphamide, auranofin, aurothioglucose, gold sodium thiomalate, penicillamine, tacrolimus or minocycline.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: NB-DMARD
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 333 | 93 | 47
NB-DMARD | 1.46 (0.67) | 1.41 (0.63) | 1.40 (0.65)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.5372, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6155, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.9696, t-test

10. Primary Outcome: Mean Number of Non-Biologic Disease Modifying Antirheumatic Drug (NB-DMARD) Received During Variable Length Pre-Index Period
Description: Mean number of NB-DMARD received during variable length pre-index period is reported. The NB-DMARD could have been hydroxychloroquine, MTX oral, leflunomide, sulfasalazine, chloroquine, cyclosporine, thalidomide, azathioprine, cyclophosphamide, auranofin, aurothioglucose, gold sodium thiomalate, penicillamine, tacrolimus or minocycline. Variable-length pre-index period defined as the period from the participant's first date of enrollment in the database to the day before the index date. The date of enrollment had to be at least 1 year prior to the index date and depending on the participant could have been as much as maximum of 5.2 years. The index date was the date of the first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During variable length pre-index period (1 year before the index date up to 5.2 years)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: NB-DMARD
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 334 | 94 | 48
NB-DMARD | 1.62 (0.77) | 1.52 (0.70) | 1.63 (0.82)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.2514, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.9851, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4309, t-test

11. Primary Outcome: Mean Quan-Charlson Comorbidity Score of Participants
Description: The mean Quan-Charlson Comorbidity Score during the Pre-Index Period is reported. Quan-Charlson Comorbidity Score predicts the probability of death within one year in participants and was based on the presence of any diagnosis codes on medical claims at any time during the 12-month pre-index period, based on the International Classification of Diseases (ICD) diagnosis codes. Total score ranges from 0 to 9.0. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome could result in mortality or higher healthcare resource utilization.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
score on a scale | 1.69 (1.08) | 1.76 (1.18) | 1.90 (1.46)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.6033, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3480, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.5375, t-test

12. Primary Outcome: Number of Participants With Top 25 Comorbid Conditions as Per Agency for Healthcare Research and Quality (AHRQ) During Pre-Index Period
Description: Top 25 comorbid conditions: 1) rheumatoid arthritis/related disease, 2)other aftercare, 3)other connective tissue disease, 4)other non-traumatic joint disorders, 5)medical examination/evaluation, 6) other suspected conditions(other miscellaneous conditions other than mental disorders/infectious disease), 7)immunizations/screening for infectious disease, 8)osteoarthritis, 9)essential hypertension, 10) residual codes: unclassified, 11)disorders of lipid metabolism, 12)back problems, 13)other upper respiratory infections, 14)other lower respiratory disease, 15)other nervous system disorders, 16)other skin disorders, 17)thyroid disorders, 18)other bone disease/musculoskeletal deformities, 19) malaise/fatigue, 20)esophageal disorders, 21)nutritional deficiencies, 22)other nutritional: endocrine, metabolic disorders, 23)diabetes mellitus without complication, 24)other/unspecified benign neoplasm, 25)genitourinary symptoms/ill-defined conditions. A participant could have had >=1 comorbidity.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study. p-value could not be calculated between reporting groups for specified rows with 100% response.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  Rheumatoid arthritis/related disease | 337 | 94 | 48
  Other aftercare | 277 | 68 | 36
  Other connective tissue disease | 203 | 66 | 26
  Other non-traumatic joint disorders | 200 | 56 | 29
  Medical examination/evaluation | 195 | 56 | 24
  Other suspected conditions | 179 | 49 | 21
  Immunizations/screening for infectious disease | 176 | 44 | 19
  Osteoarthritis | 154 | 37 | 28
  Essential hypertension | 144 | 44 | 27
  Residual codes; unclassified | 144 | 42 | 23
  Disorders of lipid metabolism | 147 | 36 | 22
  Back problems | 128 | 48 | 21
  Other upper respiratory infections | 114 | 31 | 13
  Other lower respiratory disease | 101 | 30 | 18
  Other nervous system disorders | 98 | 33 | 14
  Other skin disorders | 97 | 16 | 16
  Thyroid disorders | 95 | 24 | 9
  Other bone disease/musculoskeletal deformities | 88 | 26 | 12
  Malaise/fatigue | 81 | 21 | 9
  Esophageal disorders | 74 | 23 | 12
  Nutritional deficiencies | 75 | 22 | 12
  Other nutritional: endocrine, metabolic disorders | 74 | 17 | 12
  Diabetes mellitus without complication | 72 | 18 | 11
  Other/unspecified benign neoplasm | 65 | 18 | 5
  Genitourinary symptoms/ill-defined conditions | 59 | 12 | 9
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other aftercare; Test type: Superiority; p = 0.0345, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other aftercare; Test type: Superiority; p = 0.2316, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other aftercare; Test type: Superiority; p = 0.7349, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other connective tissue disease; Test type: Superiority; p = 0.0774, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other connective tissue disease; Test type: Superiority; p = 0.4228, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other connective tissue disease; Test type: Superiority; p = 0.0583, Chi-squared
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other non-traumatic joint disorders; Test type: Superiority; p = 0.9683, Chi-squared
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other non-traumatic joint disorders; Test type: Superiority; p = 0.8877, Chi-squared
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other non-traumatic joint disorders; Test type: Superiority; p = 0.9228, Chi-squared
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Medical examination/evaluation; Test type: Superiority; p = 0.7661, Chi-squared
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Medical examination/evaluation; Test type: Superiority; p = 0.3034, Chi-squared
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Medical examination/evaluation; Test type: Superiority; p = 0.2765, Chi-squared
Statistical Analysis 13: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other suspected conditions; Test type: Superiority; p = 0.8652, Chi-squared
Statistical Analysis 14: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other suspected conditions; Test type: Superiority; p = 0.2243, Chi-squared
Statistical Analysis 15: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other suspected conditions; Test type: Superiority; p = 0.3449, Chi-squared
Statistical Analysis 16: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Immunizations/screening for infectious disease; Test type: Superiority; p = 0.3529, Chi-squared
Statistical Analysis 17: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Immunizations/screening for infectious disease; Test type: Superiority; p = 0.1012, Chi-squared
Statistical Analysis 18: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Immunizations/screening for infectious disease; Test type: Superiority; p = 0.4123, Chi-squared
Statistical Analysis 19: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Osteoarthritis; Test type: Superiority; p = 0.2742, Chi-squared
Statistical Analysis 20: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Osteoarthritis; Test type: Superiority; p = 0.1009, Chi-squared
Statistical Analysis 21: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Osteoarthritis; Test type: Superiority; p = 0.0318, Chi-squared
Statistical Analysis 22: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Essential hypertension; Test type: Superiority; p = 0.4808, Chi-squared
Statistical Analysis 23: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Essential hypertension; Test type: Superiority; p = 0.0778, Chi-squared
Statistical Analysis 24: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Essential hypertension; Test type: Superiority; p = 0.2871, Chi-squared
Statistical Analysis 25: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Residual codes; unclassified; Test type: Superiority; p = 0.7356, Chi-squared
Statistical Analysis 26: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Residual codes; unclassified; Test type: Superiority; p = 0.4975, Chi-squared
Statistical Analysis 27: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Residual codes; unclassified; Test type: Superiority; p = 0.7143, Chi-squared
Statistical Analysis 28: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Disorders of lipid metabolism; Test type: Superiority; p = 0.3559, Chi-squared
Statistical Analysis 29: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Disorders of lipid metabolism; Test type: Superiority; p = 0.7725, Chi-squared
Statistical Analysis 30: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Disorders of lipid metabolism; Test type: Superiority; p = 0.3875, Chi-squared
Statistical Analysis 31: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Back problems; Test type: Superiority; p = 0.0225, Chi-squared
Statistical Analysis 32: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Back problems; Test type: Superiority; p = 0.4427, Chi-squared
Statistical Analysis 33: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Back problems; Test type: Superiority; p = 0.4094, Chi-squared
Statistical Analysis 34: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other upper respiratory infections; Test type: Superiority; p = 0.8775, Chi-squared
Statistical Analysis 35: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other upper respiratory infections; Test type: Superiority; p = 0.3525, Chi-squared
Statistical Analysis 36: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other upper respiratory infections; Test type: Superiority; p = 0.4724, Chi-squared
Statistical Analysis 37: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other lower respiratory disease; Test type: Superiority; p = 0.7170, Chi-squared
Statistical Analysis 38: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other lower respiratory disease; Test type: Superiority; p = 0.2909, Chi-squared
Statistical Analysis 39: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other lower respiratory disease; Test type: Superiority; p = 0.5057, Chi-squared
Statistical Analysis 40: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other nervous system disorders; Test type: Superiority; p = 0.2613, Chi-squared
Statistical Analysis 41: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nervous system disorders; Test type: Superiority; p = 0.9901, Chi-squared
Statistical Analysis 42: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nervous system disorders; Test type: Superiority; p = 0.4768, Chi-squared
Statistical Analysis 43: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other skin disorders; Test type: Superiority; p = 0.0219, Chi-squared
Statistical Analysis 44: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other skin disorders; Test type: Superiority; p = 0.5172, Chi-squared
Statistical Analysis 45: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other skin disorders; Test type: Superiority; p = 0.0278, Chi-squared
Statistical Analysis 46: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Thyroid disorders; Test type: Superiority; p = 0.6103, Chi-squared
Statistical Analysis 47: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Thyroid disorders; Test type: Superiority; p = 0.1682, Chi-squared
Statistical Analysis 48: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Thyroid disorders; Test type: Superiority; p = 0.3654, Chi-squared
Statistical Analysis 49: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other bone disease/musculoskeletal deformities; Test type: Superiority; p = 0.7637, Chi-squared
Statistical Analysis 50: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other bone disease/musculoskeletal deformities; Test type: Superiority; p = 0.8693, Chi-squared
Statistical Analysis 51: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other bone disease/musculoskeletal deformities; Test type: Superiority; p = 0.7349, Chi-squared
Statistical Analysis 52: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Malaise/fatigue; Test type: Superiority; p = 0.7324, Chi-squared
Statistical Analysis 53: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Malaise/fatigue; Test type: Superiority; p = 0.4182, Chi-squared
Statistical Analysis 54: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Malaise/fatigue; Test type: Superiority; p = 0.6200, Chi-squared
Statistical Analysis 55: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Esophageal disorders; Test type: Superiority; p = 0.6064, Chi-squared
Statistical Analysis 56: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Esophageal disorders; Test type: Superiority; p = 0.6360, Chi-squared
Statistical Analysis 57: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Esophageal disorders; Test type: Superiority; p = 0.9445, Chi-squared
Statistical Analysis 58: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Nutritional deficiencies; Test type: Superiority; p = 0.8135, Chi-squared
Statistical Analysis 59: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Nutritional deficiencies; Test type: Superiority; p = 0.6705, Chi-squared
Statistical Analysis 60: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Nutritional deficiencies; Test type: Superiority; p = 0.8331, Chi-squared
Statistical Analysis 61: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other nutritional; endocrine; and metabolic disorders; Test type: Superiority; p = 0.4158, Chi-squared
Statistical Analysis 62: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nutritional; endocrine; and metabolic disorders; Test type: Superiority; p = 0.6360, Chi-squared
Statistical Analysis 63: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nutritional; endocrine; and metabolic disorders; Test type: Superiority; p = 0.3336, Chi-squared
Statistical Analysis 64: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Diabetes mellitus without complication; Test type: Superiority; p = 0.6402, Chi-squared
Statistical Analysis 65: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diabetes mellitus without complication; Test type: Superiority; p = 0.8068, Chi-squared
Statistical Analysis 66: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diabetes mellitus without complication; Test type: Superiority; p = 0.5983, Chi-squared
Statistical Analysis 67: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other/unspecified benign neoplasm; Test type: Superiority; p = 0.9759, Chi-squared
Statistical Analysis 68: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other/unspecified benign neoplasm; Test type: Superiority; p = 0.1360, Chi-squared
Statistical Analysis 69: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other/unspecified benign neoplasm; Test type: Superiority; p = 0.1815, Chi-squared
Statistical Analysis 70: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Genitourinary symptoms/ill-defined conditions; Test type: Superiority; p = 0.2731, Chi-squared
Statistical Analysis 71: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Genitourinary symptoms/ill-defined conditions; Test type: Superiority; p = 0.8327, Chi-squared
Statistical Analysis 72: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Genitourinary symptoms/ill-defined conditions; Test type: Superiority; p = 0.3420, Chi-squared

13. Primary Outcome: Number of Participants With Top 25 Comorbid Conditions as Per Agency for Healthcare Research and Quality (AHRQ) During Post-Index Period
Description: Top 25 comorbid conditions: 1) rheumatoid arthritis/related disease, 2)other aftercare, 3)other connective tissue disease, 4)other non-traumatic joint disorders, 5)medical examination/evaluation, 6) other suspected conditions(other miscellaneous conditions other than mental disorders/infectious disease), 7)immunizations/screening for infectious disease, 8)osteoarthritis, 9)essential hypertension, 10) residual codes: unclassified, 11)disorders of lipid metabolism, 12)back problems, 13)other upper respiratory infections, 14)other lower respiratory disease, 15)other nervous system disorders, 16)other skin disorders, 17)thyroid disorders, 18)other bone disease/musculoskeletal deformities, 19) malaise/fatigue, 20)esophageal disorders, 21)nutritional deficiencies, 22)other nutritional: endocrine, metabolic disorders, 23)diabetes mellitus without complication, 24)other/unspecified benign neoplasm, 25)Other upper respiratory disease. A participant could have had >=1 comorbidity.
Time Frame: During post-index period (12 months duration post index date [Index date: date of first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years])
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  Rheumatoid arthritis/related disease | 336 | 92 | 48
  Other aftercare | 290 | 69 | 39
  Other connective tissue disease | 187 | 54 | 32
  Other suspected conditions | 186 | 57 | 29
  Medical examination/evaluation | 186 | 51 | 22
  Other non-traumatic joint disorders | 169 | 53 | 29
  Essential hypertension | 156 | 51 | 26
  Residual codes; unclassified | 165 | 42 | 23
  Disorders of lipid metabolism | 155 | 42 | 20
  Osteoarthritis | 141 | 41 | 21
  Immunizations/screening for infectious disease | 142 | 44 | 15
  Back problems | 138 | 38 | 25
  Other upper respiratory infections | 123 | 29 | 21
  Other nervous system disorders | 100 | 37 | 20
  Other lower respiratory disease | 106 | 28 | 20
  Other skin disorders | 100 | 30 | 17
  Other nutritional, endocrine, metabolic disorders | 104 | 25 | 14
  Thyroid disorders | 90 | 23 | 11
  Other bone disease/musculoskeletal deformities | 90 | 20 | 13
  Nutritional deficiencies | 74 | 25 | 16
  Diabetes mellitus without complication | 71 | 24 | 11
  Esophageal disorders | 71 | 19 | 11
  Malaise/fatigue | 69 | 17 | 7
  Other/unspecified benign neoplasm | 60 | 19 | 11
  Other upper respiratory disease | 67 | 18 | 7
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Rheumatoid arthritis/related disease; Test type: Superiority; p = 0.0590, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Rheumatoid arthritis/related disease; Test type: Superiority; p = 0.7055, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Rheumatoid arthritis/related disease; Test type: Superiority; p = 0.3088, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other aftercare; Test type: Superiority; p = 0.0036, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other aftercare; Test type: Superiority; p = 0.3772, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other aftercare; Test type: Superiority; p = 0.3000, Chi-squared
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other connective tissue disease; Test type: Superiority; p = 0.7354, Chi-squared
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other connective tissue disease; Test type: Superiority; p = 0.1435, Chi-squared
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other connective tissue disease; Test type: Superiority; p = 0.2876, Chi-squared
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other non-traumatic joint disorders; Test type: Superiority; p = 0.2848, Chi-squared
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other non-traumatic joint disorders; Test type: Superiority; p = 0.1830, Chi-squared
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other non-traumatic joint disorders; Test type: Superiority; p = 0.6453, Chi-squared
Statistical Analysis 13: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Medical examination/evaluation; Test type: Superiority; p = 0.8717, Chi-squared
Statistical Analysis 14: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Medical examination/evaluation; Test type: Superiority; p = 0.8717, Chi-squared
Statistical Analysis 15: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Medical examination/evaluation; Test type: Superiority; p = 0.3422, Chi-squared
Statistical Analysis 16: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other suspected conditions; Test type: Superiority; p = 0.3465, Chi-squared
Statistical Analysis 17: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other suspected conditions; Test type: Superiority; p = 0.4953, Chi-squared
Statistical Analysis 18: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other suspected conditions; Test type: Superiority; p = 0.9796, Chi-squared
Statistical Analysis 19: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Immunizations/screening for infectious disease; Test type: Superiority; p = 0.4187, Chi-squared
Statistical Analysis 20: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Immunizations/screening for infectious disease; Test type: Superiority; p = 0.1510, Chi-squared
Statistical Analysis 21: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Immunizations/screening for infectious disease; Test type: Superiority; p = 0.0751, Chi-squared
Statistical Analysis 22: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Osteoarthritis; Test type: Superiority; p = 0.7577, Chi-squared
Statistical Analysis 23: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Osteoarthritis; Test type: Superiority; p = 0.8020, Chi-squared
Statistical Analysis 24: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Osteoarthritis; Test type: Superiority; p = 0.9879, Chi-squared
Statistical Analysis 25: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Essential hypertension; Test type: Superiority; p = 0.1717, Chi-squared
Statistical Analysis 26: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Essential hypertension; Test type: Superiority; p = 0.3065, Chi-squared
Statistical Analysis 27: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Essential hypertension; Test type: Superiority; p = 0.9920, Chi-squared
Statistical Analysis 28: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Residual codes; unclassified; Test type: Superiority; p = 0.4626, Chi-squared
Statistical Analysis 29: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Residual codes; unclassified; Test type: Superiority; p = 0.8922, Chi-squared
Statistical Analysis 30: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Residual codes; unclassified; Test type: Superiority; p = 0.7143, Chi-squared
Statistical Analysis 31: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Disorders of lipid metabolism; Test type: Superiority; p = 0.8212, Chi-squared
Statistical Analysis 32: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Disorders of lipid metabolism; Test type: Superiority; p = 0.5732, Chi-squared
Statistical Analysis 33: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Disorders of lipid metabolism; Test type: Superiority; p = 0.7319, Chi-squared
Statistical Analysis 34: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Back problems; Test type: Superiority; p = 0.9272, Chi-squared
Statistical Analysis 35: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Back problems; Test type: Superiority; p = 0.1441, Chi-squared
Statistical Analysis 36: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Back problems; Test type: Superiority; p = 0.1859, Chi-squared
Statistical Analysis 37: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other upper respiratory infections; Test type: Superiority; p = 0.3109, Chi-squared
Statistical Analysis 38: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other upper respiratory infections; Test type: Superiority; p = 0.3313, Chi-squared
Statistical Analysis 39: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other upper respiratory infections; Test type: Superiority; p = 0.1279, Chi-squared
Statistical Analysis 40: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other lower respiratory disease; Test type: Superiority; p = 0.7575, Chi-squared
Statistical Analysis 41: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other lower respiratory disease; Test type: Superiority; p = 0.1583, Chi-squared
Statistical Analysis 42: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other lower respiratory disease; Test type: Superiority; p = 0.1569, Chi-squared
Statistical Analysis 43: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other nervous system disorders; Test type: Superiority; p = 0.0745, Chi-squared
Statistical Analysis 44: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nervous system disorders; Test type: Superiority; p = 0.0933, Chi-squared
Statistical Analysis 45: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nervous system disorders; Test type: Superiority; p = 0.7910, Chi-squared
Statistical Analysis 46: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other skin disorders; Test type: Superiority; p = 0.6755, Chi-squared
Statistical Analysis 47: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other skin disorders; Test type: Superiority; p = 0.4183, Chi-squared
Statistical Analysis 48: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other skin disorders; Test type: Superiority; p = 0.6749, Chi-squared
Statistical Analysis 49: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Thyroid disorders; Test type: Superiority; p = 0.6626, Chi-squared
Statistical Analysis 50: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Thyroid disorders; Test type: Superiority; p = 0.5766, Chi-squared
Statistical Analysis 51: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Thyroid disorders; Test type: Superiority; p = 0.8376, Chi-squared
Statistical Analysis 52: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other bone disease/musculoskeletal deformities; Test type: Superiority; p = 0.2857, Chi-squared
Statistical Analysis 53: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other bone disease/musculoskeletal deformities; Test type: Superiority; p = 0.9560, Chi-squared
Statistical Analysis 54: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other bone disease/musculoskeletal deformities; Test type: Superiority; p = 0.4384, Chi-squared
Statistical Analysis 55: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Malaise/fatigue; Test type: Superiority; p = 0.6082, Chi-squared
Statistical Analysis 56: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Malaise/fatigue; Test type: Superiority; p = 0.3374, Chi-squared
Statistical Analysis 57: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Malaise/fatigue; Test type: Superiority; p = 0.5984, Chi-squared
Statistical Analysis 58: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Esophageal disorders; Test type: Superiority; p = 0.8568, Chi-squared
Statistical Analysis 59: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Esophageal disorders; Test type: Superiority; p = 0.7698, Chi-squared
Statistical Analysis 60: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Esophageal disorders; Test type: Superiority; p = 0.7089, Chi-squared
Statistical Analysis 61: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Nutritional deficiencies; Test type: Superiority; p = 0.3446, Chi-squared
Statistical Analysis 62: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Nutritional deficiencies; Test type: Superiority; p = 0.0815, Chi-squared
Statistical Analysis 63: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Nutritional deficiencies; Test type: Superiority; p = 0.4020, Chi-squared
Statistical Analysis 64: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other nutritional: endocrine/metabolic disorders; Test type: Superiority; p = 0.4246, Chi-squared
Statistical Analysis 65: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nutritional: endocrine/metabolic disorders; Test type: Superiority; p = 0.8118, Chi-squared
Statistical Analysis 66: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other nutritional: endocrine/metabolic disorders; Test type: Superiority; p = 0.7454, Chi-squared
Statistical Analysis 67: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diabetes mellitus without complication; Test type: Superiority; p = 0.3559, Chi-squared
Statistical Analysis 68: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diabetes mellitus without complication; Test type: Superiority; p = 0.7698, Chi-squared
Statistical Analysis 69: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diabetes mellitus without complication; Test type: Superiority; p = 0.7323, Chi-squared
Statistical Analysis 70: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other/unspecified benign neoplasm; Test type: Superiority; p = 0.5935, Chi-squared
Statistical Analysis 71: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other/unspecified benign neoplasm; Test type: Superiority; p = 0.3928, Chi-squared
Statistical Analysis 72: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other/unspecified benign neoplasm; Test type: Superiority; p = 0.7089, Chi-squared
Statistical Analysis 73: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Other upper respiratory disease; Test type: Superiority; p = 0.8746, Chi-squared
Statistical Analysis 74: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other upper respiratory disease; Test type: Superiority; p = 0.3835, Chi-squared
Statistical Analysis 75: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Other upper respiratory disease; Test type: Superiority; p = 0.4992, Chi-squared

14. Primary Outcome: Mean Claims Based Index of RA Severity (CIRAS) Score During Pre-Index Period
Description: The mean of the CIRAS score during pre-index period is reported. The CIRAS is based on claims at any time during the 12-month pre-index period, used to measure RA disease severity using 9 measures (age at index, gender, inflammatory marker test ordered, rehabilitation visit, rheumatoid factor test, Felty's syndrome, number of platelet counts ordered, number of chemistry panels ordered, rheumatologist visit). Value of all 9 measure was used to derive the overall CIRAS score which ranges from 0-7.9 with higher value indicating greater severity of RA.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
score on a scale | 4.57 (1.37) | 4.76 (1.50) | 4.31 (1.20)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.2336, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2109, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0691, t-test

15. Primary Outcome: Number of Participants With 25 Most Common Medications Use During Pre-Index Period
Description: Number of participants with 25 most common medications use during the pre-index period are reported. The 25 most medications: 1) MTX sodium, 2) folic acid, 3) prednisone, 4) acetaminophen/hydrocodone bitartrate, 5) azithromycin, 6) adalimumab, 7) hydroxychloroquine sulfate, 8) etanercept, 9) levothyroxine sodium, 10) methylprednisolone, 11) omeprazole, 12) tramadol hydrochloride, 13) meloxicam, 14) amoxicillin, 15) albuterol sulfate, 16) gabapentin, 17) acetaminophen/oxycodone hydrochloride, 18) amoxicillin/clavulanate potassium, 19) cyclobenzaprine hydrochloride, 20) fluticasone propionate, 21) ciprofloxacin hydrochloride, 22) duloxetine hydrochloride, 23) atorvastatin calcium, 24) diclofenac sodium, 25) levofloxacin. A participant could have received >=1 most common medication.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  MTX Sodium | 330 | 92 | 47
  Folic Acid | 243 | 65 | 34
  Prednisone | 214 | 70 | 38
  Acetaminophen/Hydrocodone Bitartrate | 111 | 33 | 14
  Azithromycin | 80 | 28 | 15
  Adalimumab | 84 | 26 | 6
  Hydroxychloroquine Sulfate | 83 | 21 | 10
  Etanercept | 76 | 21 | 16
  Levothyroxine Sodium | 80 | 16 | 10
  Methylprednisolone | 66 | 22 | 15
  Omeprazole | 69 | 16 | 10
  Tramadol Hydrochloride | 59 | 22 | 11
  Meloxicam | 58 | 20 | 8
  Amoxicillin | 54 | 17 | 9
  Albuterol Sulfate | 58 | 17 | 4
  Gabapentin | 52 | 15 | 7
  Acetaminophen/Oxycodone Hydrochloride | 46 | 20 | 7
  Amoxicillin/Clavulanate Potassium | 53 | 11 | 6
  Cyclobenzaprine Hydrochloride | 45 | 16 | 7
  Fluticasone Propionate | 47 | 13 | 5
  Ciprofloxacin Hydrochloride | 46 | 10 | 8
  Duloxetine Hydrochloride | 42 | 17 | 4
  Atorvastatin Calcium | 44 | 11 | 7
  Diclofenac Sodium | 39 | 16 | 4
  Levofloxacin | 40 | 13 | 4
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; MTX Sodium; Test type: Superiority; p = 0.9758, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; MTX Sodium; Test type: Superiority; p = 0.9978, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; MTX Sodium; Test type: Superiority; p = 0.9861, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Folic Acid; Test type: Superiority; p = 0.5744, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Folic Acid; Test type: Superiority; p = 0.8542, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Folic Acid; Test type: Superiority; p = 0.8363, Chi-squared
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Prednisone; Test type: Superiority; p = 0.0473, Chi-squared
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Prednisone; Test type: Superiority; p = 0.0327, Chi-squared
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Prednisone; Test type: Superiority; p = 0.5348, Chi-squared
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Acetaminophen/Hydrocodone Bitartrate; Test type: Superiority; p = 0.6934, Chi-squared
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Hydrocodone Bitartrate; Test type: Superiority; p = 0.6017, Chi-squared
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Hydrocodone Bitartrate; Test type: Superiority; p = 0.4768, Chi-squared
Statistical Analysis 13: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Azithromycin; Test type: Superiority; p = 0.2315, Chi-squared
Statistical Analysis 14: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Azithromycin; Test type: Superiority; p = 0.2588, Chi-squared
Statistical Analysis 15: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Azithromycin; Test type: Superiority; p = 0.8576, Chi-squared
Statistical Analysis 16: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Adalimumab; Test type: Superiority; p = 0.5909, Chi-squared
Statistical Analysis 17: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Adalimumab; Test type: Superiority; p = 0.0570, Chi-squared
Statistical Analysis 18: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Adalimumab; Test type: Superiority; p = 0.0408, Chi-squared
Statistical Analysis 19: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Hydroxychloroquine Sulfate; Test type: Superiority; p = 0.6465, Chi-squared
Statistical Analysis 20: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Hydroxychloroquine Sulfate; Test type: Superiority; p = 0.5654, Chi-squared
Statistical Analysis 21: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Hydroxychloroquine Sulfate; Test type: Superiority; p = 0.8371, Chi-squared
Statistical Analysis 22: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Etanercept; Test type: Superiority; p = 0.9654, Chi-squared
Statistical Analysis 23: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Etanercept; Test type: Superiority; p = 0.1013, Chi-squared
Statistical Analysis 24: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Etanercept; Test type: Superiority; p = 0.1580, Chi-squared
Statistical Analysis 25: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Levothyroxine Sodium; Test type: Superiority; p = 0.1663, Chi-squared
Statistical Analysis 26: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levothyroxine Sodium; Test type: Superiority; p = 0.6563, Chi-squared
Statistical Analysis 27: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levothyroxine Sodium; Test type: Superiority; p = 0.5785, Chi-squared
Statistical Analysis 28: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Methylprednisolone; Test type: Superiority; p = 0.4166, Chi-squared
Statistical Analysis 29: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Methylprednisolone; Test type: Superiority; p = 0.0636, Chi-squared
Statistical Analysis 30: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Methylprednisolone; Test type: Superiority; p = 0.3137, Chi-squared
Statistical Analysis 31: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Omeprazole; Test type: Superiority; p = 0.4568, Chi-squared
Statistical Analysis 32: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Omeprazole; Test type: Superiority; p = 0.5785, Chi-squared
Statistical Analysis 33: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Omeprazole; Test type: Superiority; p = 0.9541, Chi-squared
Statistical Analysis 34: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Tramadol Hydrochloride; Test type: Superiority; p = 0.1956, Chi-squared
Statistical Analysis 35: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Tramadol Hydrochloride; Test type: Superiority; p = 0.3633, Chi-squared
Statistical Analysis 36: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Tramadol Hydrochloride; Test type: Superiority; p = 0.9481, Chi-squared
Statistical Analysis 37: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Meloxicam; Test type: Superiority; p = 0.3653, Chi-squared
Statistical Analysis 38: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Meloxicam; Test type: Superiority; p = 0.9255, Chi-squared
Statistical Analysis 39: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Meloxicam; Test type: Superiority; p = 0.5137, Chi-squared
Statistical Analysis 40: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Amoxicillin; Test type: Superiority; p = 0.6338, Chi-squared
Statistical Analysis 41: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin; Test type: Superiority; p = 0.6329, Chi-squared
Statistical Analysis 42: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin; Test type: Superiority; p = 0.9228, Chi-squared
Statistical Analysis 43: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Albuterol Sulfate; Test type: Superiority; p = 0.8433, Chi-squared
Statistical Analysis 44: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Albuterol Sulfate; Test type: Superiority; p = 0.1175, Chi-squared
Statistical Analysis 45: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Albuterol Sulfate; Test type: Superiority; p = 0.1215, Chi-squared
Statistical Analysis 46: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Gabapentin; Test type: Superiority; p = 0.9007, Chi-squared
Statistical Analysis 47: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Gabapentin; Test type: Superiority; p = 0.8789, Chi-squared
Statistical Analysis 48: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Gabapentin; Test type: Superiority; p = 0.8305, Chi-squared
Statistical Analysis 49: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Acetaminophen/Oxycodone Hydrochloride; Test type: Superiority; p = 0.0694, Chi-squared
Statistical Analysis 50: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Oxycodone Hydrochloride; Test type: Superiority; p = 0.8606, Chi-squared
Statistical Analysis 51: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Oxycodone Hydrochloride; Test type: Superiority; p = 0.3363, Chi-squared
Statistical Analysis 52: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Amoxicillin/Clavulanate Potassium; Test type: Superiority; p = 0.3319, Chi-squared
Statistical Analysis 53: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin/Clavulanate Potassium; Test type: Superiority; p = 0.5615, Chi-squared
Statistical Analysis 54: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin/Clavulanate Potassium; Test type: Superiority; p = 0.8898, Chi-squared
Statistical Analysis 55: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Cyclobenzaprine Hydrochloride; Test type: Superiority; p = 0.3670, Chi-squared
Statistical Analysis 56: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cyclobenzaprine Hydrochloride; Test type: Superiority; p = 0.8155, Chi-squared
Statistical Analysis 57: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cyclobenzaprine Hydrochloride; Test type: Superiority; p = 0.7091, Chi-squared
Statistical Analysis 58: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Fluticasone Propionate; Test type: Superiority; p = 0.9769, Chi-squared
Statistical Analysis 59: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Fluticasone Propionate; Test type: Superiority; p = 0.5032, Chi-squared
Statistical Analysis 60: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Fluticasone Propionate; Test type: Superiority; p = 0.5631, Chi-squared
Statistical Analysis 61: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Ciprofloxacin Hydrochloride; Test type: Superiority; p = 0.4426, Chi-squared
Statistical Analysis 62: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Ciprofloxacin Hydrochloride; Test type: Superiority; p = 0.5734, Chi-squared
Statistical Analysis 63: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Ciprofloxacin Hydrochloride; Test type: Superiority; p = 0.3071, Chi-squared
Statistical Analysis 64: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Duloxetine Hydrochloride; Test type: Superiority; p = 0.1608, Chi-squared
Statistical Analysis 65: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Duloxetine Hydrochloride; Test type: Superiority; p = 0.4092, Chi-squared
Statistical Analysis 66: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Duloxetine Hydrochloride; Test type: Superiority; p = 0.1215, Chi-squared
Statistical Analysis 67: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Atorvastatin Calcium; Test type: Superiority; p = 0.7279, Chi-squared
Statistical Analysis 68: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Atorvastatin Calcium; Test type: Superiority; p = 0.7703, Chi-squared
Statistical Analysis 69: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Atorvastatin Calcium; Test type: Superiority; p = 0.6254, Chi-squared
Statistical Analysis 70: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Diclofenac Sodium; Test type: Superiority; p = 0.1615, Chi-squared
Statistical Analysis 71: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diclofenac Sodium; Test type: Superiority; p = 0.5050, Chi-squared
Statistical Analysis 72: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diclofenac Sodium; Test type: Superiority; p = 0.1592, Chi-squared
Statistical Analysis 73: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Levofloxacin; Test type: Superiority; p = 0.6088, Chi-squared
Statistical Analysis 74: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levofloxacin; Test type: Superiority; p = 0.4713, Chi-squared
Statistical Analysis 75: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levofloxacin; Test type: Superiority; p = 0.3399, Chi-squared

16. Primary Outcome: Number of Participants With 26 Most Common Medications Use During Post-Index Period
Description: Number of participants with 26 most common medications use during the post-index period are reported. The 26 most common medications: 1) MTX sodium, 2) folic acid, 3) prednisone, 4) acetaminophen/hydrocodone bitartrate, 5) azithromycin, 6) adalimumab, 7) hydroxychloroquine sulfate, 8) etanercept, 9) levothyroxine sodium, 10) methylprednisolone, 11) omeprazole, 12) tramadol hydrochloride, 13) meloxicam, 14) amoxicillin, 15) albuterol sulfate, 16) gabapentin, 17) acetaminophen/oxycodone hydrochloride, 18) amoxicillin/clavulanate potassium, 19) cyclobenzaprine hydrochloride, 20) fluticasone propionate, 21) ciprofloxacin hydrochloride, 22) duloxetine hydrochloride, 23) diclofenac Sodium, 24) levofloxacin, 25) cephalexin, 26) ibuprofen. A participant could have received >=1 most common medication.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  MTX Sodium | 332 | 94 | 48
  Folic Acid | 254 | 68 | 35
  Prednisone | 260 | 81 | 43
  Acetaminophen/Hydrocodone Bitartrate | 184 | 58 | 23
  Azithromycin | 153 | 47 | 25
  Adalimumab | 126 | 37 | 11
  Hydroxychloroquine Sulfate | 108 | 25 | 13
  Etanercept | 112 | 27 | 17
  Levothyroxine Sodium | 82 | 16 | 10
  Methylprednisolone | 123 | 43 | 22
  Omeprazole | 89 | 20 | 13
  Tramadol Hydrochloride | 96 | 39 | 17
  Meloxicam | 96 | 25 | 10
  Amoxicillin | 105 | 28 | 15
  Albuterol Sulfate | 91 | 25 | 8
  Gabapentin | 78 | 21 | 11
  Acetaminophen/Oxycodone Hydrochloride | 80 | 30 | 15
  Amoxicillin/Clavulanate Potassium | 94 | 20 | 14
  Cyclobenzaprine Hydrochloride | 83 | 31 | 11
  Fluticasone Propionate | 83 | 24 | 13
  Ciprofloxacin Hydrochloride | 88 | 26 | 11
  Duloxetine Hydrochloride | 52 | 23 | 8
  Diclofenac Sodium | 71 | 27 | 10
  Levofloxacin | 79 | 24 | 12
  Cephalexin | 76 | 15 | 11
  Ibuprofen | 50 | 22 | 11
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; MTX Sodium; Test type: Superiority; p = 0.2349, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; MTX Sodium; Test type: Superiority; p = 0.3956, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Folic Acid; Test type: Superiority; p = 0.5500, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Folic Acid; Test type: Superiority; p = 0.7131, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Folic Acid; Test type: Superiority; p = 0.9420, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Prednisone; Test type: Superiority; p = 0.0571, Chi-squared
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Prednisone; Test type: Superiority; p = 0.0490, Chi-squared
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Prednisone; Test type: Superiority; p = 0.5631, Chi-squared
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Acetaminophen/Hydrocodone Bitartrate; Test type: Superiority; p = 0.2198, Chi-squared
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Hydrocodone Bitartrate; Test type: Superiority; p = 0.3850, Chi-squared
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Hydrocodone Bitartrate; Test type: Superiority; p = 0.1165, Chi-squared
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Azithromycin; Test type: Superiority; p = 0.4291, Chi-squared
Statistical Analysis 13: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Azithromycin; Test type: Superiority; p = 0.3850, Chi-squared
Statistical Analysis 14: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Azithromycin; Test type: Superiority; p = 0.8143, Chi-squared
Statistical Analysis 15: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Adalimumab; Test type: Superiority; p = 0.7272, Chi-squared
Statistical Analysis 16: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Adalimumab; Test type: Superiority; p = 0.0501, Chi-squared
Statistical Analysis 17: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Adalimumab; Test type: Superiority; p = 0.0500, Chi-squared
Statistical Analysis 18: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Hydroxychloroquine Sulfate; Test type: Superiority; p = 0.3116, Chi-squared
Statistical Analysis 19: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Hydroxychloroquine Sulfate; Test type: Superiority; p = 0.4882, Chi-squared
Statistical Analysis 20: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Hydroxychloroquine Sulfate; Test type: Superiority; p = 0.9505, Chi-squared
Statistical Analysis 21: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Etanercept; Test type: Superiority; p = 0.4080, Chi-squared
Statistical Analysis 22: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Etanercept; Test type: Superiority; p = 0.7644, Chi-squared
Statistical Analysis 23: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Etanercept; Test type: Superiority; p = 0.4146, Chi-squared
Statistical Analysis 24: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Levothyroxine Sodium; Test type: Superiority; p = 0.1348, Chi-squared
Statistical Analysis 25: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levothyroxine Sodium; Test type: Superiority; p = 0.5948, Chi-squared
Statistical Analysis 26: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levothyroxine Sodium; Test type: Superiority; p = 0.5785, Chi-squared
Statistical Analysis 27: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Methylprednisolone; Test type: Superiority; p = 0.1033, Chi-squared
Statistical Analysis 28: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Methylprednisolone; Test type: Superiority; p = 0.2117, Chi-squared
Statistical Analysis 29: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Methylprednisolone; Test type: Superiority; p = 0.9920, Chi-squared
Statistical Analysis 30: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Omeprazole; Test type: Superiority; p = 0.9212, Chi-squared
Statistical Analysis 31: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Omeprazole; Test type: Superiority; p = 0.9212, Chi-squared
Statistical Analysis 32: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Omeprazole; Test type: Superiority; p = 0.4384, Chi-squared
Statistical Analysis 33: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Tramadol Hydrochloride; Test type: Superiority; p = 0.0162, Chi-squared
Statistical Analysis 34: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Tramadol Hydrochloride; Test type: Superiority; p = 0.3239, Chi-squared
Statistical Analysis 35: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Tramadol Hydrochloride; Test type: Superiority; p = 0.4837, Chi-squared
Statistical Analysis 36: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Meloxicam; Test type: Superiority; p = 0.7183, Chi-squared
Statistical Analysis 37: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Meloxicam; Test type: Superiority; p = 0.2667, Chi-squared
Statistical Analysis 38: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Meloxicam; Test type: Superiority; p = 0.4510, Chi-squared
Statistical Analysis 39: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Amoxicillin; Test type: Superiority; p = 0.7993, Chi-squared
Statistical Analysis 40: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin; Test type: Superiority; p = 0.9896, Chi-squared
Statistical Analysis 41: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin; Test type: Superiority; p = 0.8576, Chi-squared
Statistical Analysis 42: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Albuterol Sulfate; Test type: Superiority; p = 0.9373, Chi-squared
Statistical Analysis 43: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Albuterol Sulfate; Test type: Superiority; p = 0.1253, Chi-squared
Statistical Analysis 44: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Albuterol Sulfate; Test type: Superiority; p = 0.1851, Chi-squared
Statistical Analysis 45: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Gabapentin; Test type: Superiority; p = 0.8697, Chi-squared
Statistical Analysis 46: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Gabapentin; Test type: Superiority; p = 0.9719, Chi-squared
Statistical Analysis 47: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Gabapentin; Test type: Superiority; p = 0.9380, Chi-squared
Statistical Analysis 48: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Acetaminophen/Oxycodone Hydrochloride; Test type: Superiority; p = 0.1079, Chi-squared
Statistical Analysis 49: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Oxycodone Hydrochloride; Test type: Superiority; p = 0.2588, Chi-squared
Statistical Analysis 50: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Acetaminophen/Oxycodone Hydrochloride; Test type: Superiority; p = 0.9358, Chi-squared
Statistical Analysis 51: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Amoxicillin/Clavulanate Potassium; Test type: Superiority; p = 0.1984, Chi-squared
Statistical Analysis 52: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin/Clavulanate Potassium; Test type: Superiority; p = 0.8542, Chi-squared
Statistical Analysis 53: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Amoxicillin/Clavulanate Potassium; Test type: Superiority; p = 0.2973, Chi-squared
Statistical Analysis 54: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Cyclobenzaprine Hydrochloride; Test type: Superiority; p = 0.1046, Chi-squared
Statistical Analysis 55: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cyclobenzaprine Hydrochloride; Test type: Superiority; p = 0.7961, Chi-squared
Statistical Analysis 56: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cyclobenzaprine Hydrochloride; Test type: Superiority; p = 0.2140, Chi-squared
Statistical Analysis 57: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Fluticasone Propionate; Test type: Superiority; p = 0.8578, Chi-squared
Statistical Analysis 58: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Fluticasone Propionate; Test type: Superiority; p = 0.7131, Chi-squared
Statistical Analysis 59: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Fluticasone Propionate; Test type: Superiority; p = 0.8421, Chi-squared
Statistical Analysis 60: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Ciprofloxacin Hydrochloride; Test type: Superiority; p = 0.7637, Chi-squared
Statistical Analysis 61: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Ciprofloxacin Hydrochloride; Test type: Superiority; p = 0.6355, Chi-squared
Statistical Analysis 62: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Ciprofloxacin Hydrochloride; Test type: Superiority; p = 0.5425, Chi-squared
Statistical Analysis 63: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Duloxetine Hydrochloride; Test type: Superiority; p = 0.0410, Chi-squared
Statistical Analysis 64: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Duloxetine Hydrochloride; Test type: Superiority; p = 0.8251, Chi-squared
Statistical Analysis 65: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Duloxetine Hydrochloride; Test type: Superiority; p = 0.2871, Chi-squared
Statistical Analysis 66: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Diclofenac Sodium; Test type: Superiority; p = 0.1174, Chi-squared
Statistical Analysis 67: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diclofenac Sodium; Test type: Superiority; p = 0.9702, Chi-squared
Statistical Analysis 68: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diclofenac Sodium; Test type: Superiority; p = 0.3109, Chi-squared
Statistical Analysis 69: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Levofloxacin; Test type: Superiority; p = 0.6744, Chi-squared
Statistical Analysis 70: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levofloxacin; Test type: Superiority; p = 0.8121, Chi-squared
Statistical Analysis 71: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Levofloxacin; Test type: Superiority; p = 0.9451, Chi-squared
Statistical Analysis 72: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Cephalexin; Test type: Superiority; p = 0.1660, Chi-squared
Statistical Analysis 73: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cephalexin; Test type: Superiority; p = 0.9549, Chi-squared
Statistical Analysis 74: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cephalexin; Test type: Superiority; p = 0.3104, Chi-squared
Statistical Analysis 75: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Ibuprofen; Test type: Superiority; p = 0.0489, Chi-squared
Statistical Analysis 76: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Ibuprofen; Test type: Superiority; p = 0.1515, Chi-squared
Statistical Analysis 77: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Ibuprofen; Test type: Superiority; p = 0.9481, Chi-squared

17. Primary Outcome: Number of Participants Who Used Opioids During Pre-Index Period
Description: Number of participants who used at least one opioid during pre-index period are reported.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 173 | 55 | 27
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.2178, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.5237, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7964, Chi-squared

18. Primary Outcome: Number of Participants Who Used Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) During Pre-Index Period
Description: Number of participants who used at least one NSAID during pre-index period are reported.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 160 | 44 | 21
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.9085, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6283, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7293, Chi-squared

19. Primary Outcome: Number of Participants Who Used Opioids During Post-Index Period
Description: Number of participants who used at least one opioid during the post-index period are reported.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 170 | 47 | 28
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.9392, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3063, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3467, Chi-squared

20. Primary Outcome: Number of Participants Who Used NSAIDs During Post-Index Period
Description: Number of participants who used at least one NSAID during the post-index period are reported.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 152 | 41 | 24
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.7977, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.5241, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4702, Chi-squared

21. Primary Outcome: Mean Number of Pharmacy Claims for Opioids During Pre-Index Period
Description: The mean number of pharmacy claims for opioids during the pre-index period are reported. A pharmacy claim is defined as a claim made by participants to their insurance provider in purchasing opioids from their pharmacy.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study. Here, "overall number of participants analyzed" signifies the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pharmacy claims
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 173 | 55 | 27
pharmacy claims | 5.21 (5.48) | 6.83 (7.33) | 9.00 (12.29)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.1461, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1411, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4201, t-test

22. Primary Outcome: Mean Number of Pharmacy Claims for Non-Steroidal Anti Inflammatory Drugs (NSAIDs) During Pre-Index Period
Description: The mean number of pharmacy claims for NSAIDs during the pre-index period are reported. A pharmacy claim is defined as a claim made by participants to their insurance provider in purchasing NSAIDs from their pharmacy.
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: pharmacy claims
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 160 | 44 | 21
pharmacy claims | 3.81 (3.05) | 4.29 (3.68) | 3.48 (2.91)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.3955, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6356, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3833, t-test

23. Primary Outcome: Mean Number of Pharmacy Claims for Opioids During Post-Index Period
Description: The mean number of pharmacy claims for opioids during the post-index period are reported. A pharmacy claim is defined as a claim made by participants to their insurance provider in purchasing opioids from their pharmacy.
Time Frame: as for outcome 13
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: pharmacy claims
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 170 | 47 | 28
pharmacy claims | 5.35 (5.28) | 6.51 (7.57) | 7.29 (9.37)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.3292, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2959, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6962, t-test

24. Primary Outcome: Mean Number of Pharmacy Claims for Non-Steroidal Anti Inflammatory Drugs (NSAIDs) During Post-Index Period
Description: The mean number of pharmacy claims for NSAIDs during the post-index period are reported. A pharmacy claim is defined as a claim made by participants to their insurance provider in purchasing NSAIDs from their pharmacy.
Time Frame: as for outcome 13
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: pharmacy claims
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 152 | 41 | 24
pharmacy claims | 4.40 (3.83) | 4.57 (3.77) | 3.00 (1.80)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8138, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0070, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0358, t-test

25. Primary Outcome: Mean Number of Days From The Index Date to The First Opioid Claim During Post Index Period
Description: Mean number of days from the index date to the first opioid claim during post index period are reported.
Time Frame: as for outcome 13
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 170 | 47 | 28
days | 106.71 (96.40) | 109.93 (108.35) | 92.85 (81.74)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8453, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4806, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4809, t-test

26. Primary Outcome: Mean Number of Days From The Index Date to The First NSAIDs Claim During Post Index Period
Description: Mean number of days from the index date to the first NSAIDs claim during post index period are reported.
Time Frame: as for outcome 13
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 152 | 41 | 24
days | 100.25 (91.68) | 117.00 (93.12) | 124.08 (108.34)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.3076, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2509, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7827, t-test

27. Primary Outcome: Number of Participants Who Used Opioids During Tofacitinib Persistency and Post-Persistency
Description: Number of participants who used opioids during tofacitinib persistency and post-persistency are reported. Persistence for participants is defined as the period of treatment with tofacitinib. Post persistence refers to switching to another medication from tofacitinib; or discontinuing tofacitinib either permanently or for a gap in time >60 days before restarting.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  During Persistency | 159 | 40 | 25
  Post Persistency | 49 | 20 | 11
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; During Persistency; Test type: Superiority; p = 0.4261, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; During Persistency; Test type: Superiority; p = 0.5247, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; During Persistency; Test type: Superiority; p = 0.2809, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Post Persistency; Test type: Superiority; p = 0.1153, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Post Persistency; Test type: Superiority; p = 0.1344, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Post Persistency; Test type: Superiority; p = 0.8229, Chi-squared

28. Primary Outcome: Number of Participants Who Used NSAIDs During Tofacitinib Persistency and Post-Persistency
Description: Number of participants who used NSAIDs during tofacitinib persistency and post-persistency are reported. Persistence for participants is defined as the period of treatment with tofacitinib. Post persistence refers to switching to another medication from tofacitinib; or discontinuing tofacitinib either permanently or for a gap in time >60 days before restarting.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  During Persistency | 138 | 37 | 21
  Post Persistency | 51 | 17 | 8
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; During Persistency; Test type: Superiority; p = 0.7816, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; During Persistency; Test type: Superiority; p = 0.7124, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; During Persistency; Test type: Superiority; p = 0.6148, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Post Persistency; Test type: Superiority; p = 0.4876, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Post Persistency; Test type: Superiority; p = 0.7826, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Post Persistency; Test type: Superiority; p = 0.8337, Chi-squared

29. Primary Outcome: Number of Participants Who Used Oral Corticosteroids During Pre-Index Period
Description: The number of participants who used at least one oral corticosteroid during the pre-index period is reported.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 243 | 75 | 43
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.1344, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0095, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1406, Chi-squared

30. Primary Outcome: Number of Participants Who Used Oral Corticosteroids During Post-Index Period
Description: The number of participants who used at least one oral corticosteroid during the post-index period is reported.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 213 | 59 | 34
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.9379, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3025, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3388, Chi-squared

31. Primary Outcome: Mean Total Dose of Oral Corticosteroids During Pre-Index Period
Description: Mean total dose of oral corticosteroids during pre-index period is reported. The total dose is expressed as a prednisone-equivalent dose of the oral corticosteroids used.
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: milligram(mg)
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 243 | 75 | 43
milligram(mg) | 1617.82 (2148.87) | 1572.15 (1266.59) | 1209.77 (978.90)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8205, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0467, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1083, t-test

32. Primary Outcome: Mean Total Dose of Oral Corticosteroid During Post-Index Period
Description: Mean total dose of oral corticosteroids during post-index period is reported. The total dose is expressed as a prednisone-equivalent dose of the oral corticosteroids used.
Time Frame: as for outcome 13
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 213 | 59 | 34
mg | 1792.20 (3855.57) | 1871.85 (4092.22) | 1593.97 (1724.89)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8899, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6183, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6496, t-test

33. Primary Outcome: Mean Number of Visits to Rheumatologist During Pre-Index Period
Description: Mean number of visits to a rheumatologist during pre-index period is reported. A visit is referring to out-patient visit specifically to a rheumatologist.
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 259 | 74 | 34
visits | 5.43 (3.27) | 5.14 (3.50) | 4.74 (2.74)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.5027, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2375, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.5577, t-test

34. Primary Outcome: Mean Number of Visits to Rheumatologist During Variable-Length Pre-Index Period
Description: Mean number of visits to rheumatologist during the variable-length pre-index period is reported. A visit is referring to out-patient visit specifically to a rheumatologist. Variable-length pre-index period defined as the period from the participant's first date of enrollment in the database to the day before the index date. The date of enrollment had to be at least 1 year prior to the index date and depending on the participant could have been as much as maximum of 5.2 years. The index date was the date of the first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During variable length pre-index period (1 year before the index date up to 5.2 years)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 276 | 76 | 37
visits | 12.20 (9.28) | 11.72 (8.68) | 10.16 (6.22)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.6908, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0859, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2764, t-test

35. Primary Outcome: Mean Disease Duration
Description: Mean Disease Duration of RA based upon the variable length pre-index period is reported. Disease duration (in days) defined as the number of days from the earliest claim with a diagnosis of RA in the variable length pre-index period until the index date. Variable-length pre-index period defined as the period from the participant's first date of enrollment in the database to the day before the index date. The date of enrollment had to be at least 1 year prior to the index date and depending on the participant could have been as much as maximum of 5.2 years. The index date was the date of the first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During variable length pre-index period (1 year before the index date up to 5.2 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
days | 852.13 (431.04) | 786.30 (428.83) | 862.75 (462.33)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.1906, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.8744, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3295, t-test

36. Primary Outcome: Mean Out of Pocket Health Care Costs for Healthcare Services During Pre-Index Period
Description: Mean out of pocket health care costs for healthcare services during pre-index period is reported. It is categorized as: All causes and RA related. All cause consisted of money spent by participants on all health care services (pharmacy, medical [ambulatory, emergency department and inpatient admission]). RA related signifies money spent by participants on health care services for RA.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars
  All cause | 2471.36 (1952.53) | 3296.62 (2643.12) | 2233.31 (1674.19)
  RA related | 1261.49 (1578.25) | 1484.58 (1600.74) | 1002.81 (1364.90)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; All cause; Test type: Superiority; p = 0.0056, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; All cause; Test type: Superiority; p = 0.4222, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; All cause; Test type: Superiority; p = 0.0041, t-test
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; RA related; Test type: Superiority; p = 0.2277, t-test
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; RA related; Test type: Superiority; p = 0.2812, t-test
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; RA related; Test type: Superiority; p = 0.0772, t-test

37. Primary Outcome: Mean Out of Pocket Health Care Costs for Healthcare Services During Variable Length Pre-Index Period
Description: Mean out of pocket health care costs for healthcare services during variable length pre-index period is reported. It is categorized as: All causes and RA related. All cause consisted of money spent by participants on all health care services (pharmacy, medical [ambulatory, emergency department and inpatient admission]). RA related signifies one spent by participants on health care services for RA. Variable-length pre-index period defined as the period from the participant's first date of enrollment in the database to the day before the index date. The date of enrollment had to be at least 1 year prior to the index date and depending on the participant could have been as much as maximum of 5.2 years. The index date was the date of the first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During variable length pre-index period (1 year before the index date up to 5.2 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars
  All cause | 7031.96 (6241.15) | 7779.41 (5492.89) | 6451.08 (4604.24)
  RA related | 3023.26 (4459.08) | 3049.87 (2804.35) | 2684.47 (2577.28)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; All cause; Test type: Superiority; p = 0.2930, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; All cause; Test type: Superiority; p = 0.4390, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; All cause; Test type: Superiority; p = 0.1530, t-test
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; RA related; Test type: Superiority; p = 0.9439, t-test
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; RA related; Test type: Superiority; p = 0.4477, t-test
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; RA related; Test type: Superiority; p = 0.4519, t-test

38. Primary Outcome: Number of Participants With Comorbidities of Interest During Pre-Index Period
Description: Number of participants with at least one of comorbidity of interest during pre-index period is reported. The comorbidities of interest included cardiovascular diseases, chronic obstructive pulmonary disorder (COPD), asthma, kidney disease, diabetes, depression, anxiety, liver disease, sleep disorders. A participant could have >1 comorbidity of interest.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  Cardiovascular Disease | 90 | 25 | 12
  COPD | 20 | 7 | 4
  Asthma | 33 | 8 | 4
  Kidney disease | 17 | 5 | 3
  Diabetes | 58 | 16 | 8
  Depression | 44 | 12 | 6
  Anxiety | 36 | 14 | 8
  Liver disease | 13 | 2 | 3
  Sleep disorders | 43 | 13 | 10
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Cardiovascular Disease; Test type: Superiority; p = 0.9829, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cardiovascular Disease; Test type: Superiority; p = 0.8021, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Cardiovascular Disease; Test type: Superiority; p = 0.8376, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; COPD; Test type: Superiority; p = 0.5927, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; COPD; Test type: Superiority; p = 0.5202, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; COPD; Test type: Superiority; p = 0.8517, Chi-squared
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Asthma; Test type: Superiority; p = 8.33, Chi-squared
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Asthma; Test type: Superiority; p = 0.7483, Chi-squared
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Asthma; Test type: Superiority; p = 0.9713, Chi-squared
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Kidney disease; Test type: Superiority; p = 0.9148, Chi-squared
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Kidney disease; Test type: Superiority; p = 0.7248, Chi-squared
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Kidney disease; Test type: Superiority; p = 0.8200, Chi-squared
Statistical Analysis 13: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Diabetes; Test type: Superiority; p = 0.9657, Chi-squared
Statistical Analysis 14: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diabetes; Test type: Superiority; p = 0.9255, Chi-squared
Statistical Analysis 15: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Diabetes; Test type: Superiority; p = 0.9575, Chi-squared
Statistical Analysis 16: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Depression; Test type: Superiority; p = 0.9410, Chi-squared
Statistical Analysis 17: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Depression; Test type: Superiority; p = 0.9146, Chi-squared
Statistical Analysis 18: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Depression; Test type: Superiority; p = 0.9641, Chi-squared
Statistical Analysis 19: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Anxiety; Test type: Superiority; p = 0.2596, Chi-squared
Statistical Analysis 20: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Anxiety; Test type: Superiority; p = 0.2228, Chi-squared
Statistical Analysis 21: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Anxiety; Test type: Superiority; p = 0.7824, Chi-squared
Statistical Analysis 22: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Liver disease; Test type: Superiority; p = 0.4184, Chi-squared
Statistical Analysis 23: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Liver disease; Test type: Superiority; p = 0.4371, Chi-squared
Statistical Analysis 24: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Liver disease; Test type: Superiority; p = 0.2074, Chi-squared
Statistical Analysis 25: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Sleep disorders; Test type: Superiority; p = 0.7850, Chi-squared
Statistical Analysis 26: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Sleep disorders; Test type: Superiority; p = 0.1288, Chi-squared
Statistical Analysis 27: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Sleep disorders; Test type: Superiority; p = 0.2839, Chi-squared

39. Primary Outcome: Number of Participants With Non-persistence to Index Medication (Tofacitinib)
Description: Non-persistence was defined as the gap of at least 60 days in treatment with the index medication (tofacitinib) or switching to other biologic.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 110 | 37 | 27
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.2242, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0014, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0557, Chi-squared

40. Primary Outcome: Number of Participants With Post-Persistence Treatment Patterns
Description: Number of participants with post-persistence treatment patterns is reported. Post-persistence was categorized as: 1) switch immediately (if participants initiated a non-index biologic before a 60-day gap in treatment is observed for the index medication); 2) discontinue then restart (if there was a gap in the index therapy of at least 60 days and the first medication observed after the gap is the index medication); 3) discontinue then switch ( if there was a gap in the index therapy of at least 60 days and the first medication observed after the gap is a biologic [including Tofacitinib] different from index medication), 4) discontinue without switch or restart (if participant's had a gap in therapy of at least 60 days and there are no claims for either the index medication or a different biologic for the remaining observation period).
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  Switch immediately | 58 | 14 | 8
  Discontinue then switch | 6 | 3 | 3
  Discontinue then restart | 17 | 8 | 5
  Discontinue without switch or restart | 29 | 12 | 11
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Switch immediately; Test type: Superiority; p = 0.5944, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Switch immediately; Test type: Superiority; p = 0.9255, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Switch immediately; Test type: Superiority; p = 0.7824, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Discontinue then switch; Test type: Superiority; p = 0.3975, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Discontinue then switch; Test type: Superiority; p = 0.0552, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Discontinue then switch; Test type: Superiority; p = 0.3914, Chi-squared
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Discontinue then restart; Test type: Superiority; p = 0.2036, Chi-squared
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Discontinue then restart; Test type: Superiority; p = 0.1336, Chi-squared
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Discontinue then restart; Test type: Superiority; p = 0.7095, Chi-squared
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Discontinue without switch or restart; Test type: Superiority; p = 0.2241, Chi-squared
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Discontinue without switch or restart; Test type: Superiority; p = 0.0024, Chi-squared
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Discontinue without switch or restart; Test type: Superiority; p = 0.1204, Chi-squared

41. Primary Outcome: Number of Participants Who Switched From Index Medication (Tofacitinib) at Any Time During Post-Index Period
Description: Number of participants who switched from index medication (tofacitinib) to a biologic at any time during post-index period is reported.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 64 | 17 | 12
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8424, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3278, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3336, Chi-squared

42. Primary Outcome: Number of Participants Who Re-started Index Medication (Tofacitinib) at Any Time During Post-Index Period
Description: Number of participants who re-started tofacitinib (after considered as non-persistence with the tofacitinib) after discontinuation at any time during post-index period is reported.
Time Frame: as for outcome 13
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 110 | 37 | 27
Participants | 17 | 8 | 5
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.2036, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1336, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7095, Chi-squared

43. Primary Outcome: Mean Medication Possession Ratio (MPR) for Methotrexate (MTX)
Description: Mean MPR for Methotrexate is reported. MPR was calculated as the total days supply of MTX between the first and including the last prescription/administration divided by the time between the first through and including last biologic prescription/administration days supply.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study. Analysis was performed on "MTX persistent" participants only and the data for this OM was not planned to be collected and analyzed for "MTX Discontinued" and "MTX Interrupted".
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent
Number analyzed (Participants) | 337
ratio | 0.93 (0.11)

44. Primary Outcome: Mean Adherence To Methotrexate (MTX)
Description: Mean adherence for methotrexate is reported. Adherence was calculated as the total number of days supplied for MTX during the post-index period divided by the number of days from the first claim during the post-index period to the end of the post-index period
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
ratio | 0.89 (0.11) | 0.43 (0.19) | 0.58 (0.15)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p < 0.0001, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p < .0001, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p < .0001, t-test

45. Primary Outcome: Number of Participants Who Used Additional NB-DMARD During Post Index Period
Description: Number of participants who used additional NB-DMARD during post index period is reported. Additional NB-DMARD use could have been leflunomide, sulfasalazine and hydroxychloroquine.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants
  Leflunomide | 7 | 6 | 1
  Sulfasalazine | 3 | 4 | 1
  Hydroxychloroquine | 10 | 2 | 1
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Leflunomide; Test type: Superiority; p = 0.0309, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Leflunomide; Test type: Superiority; p = 0.9978, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Leflunomide; Test type: Superiority; p = 0.2629, Chi-squared
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Sulfasalazine; Test type: Superiority; p = 0.0225, Chi-squared
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Sulfasalazine; Test type: Superiority; p = 0.4456, Chi-squared
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Sulfasalazine; Test type: Superiority; p = 0.5065, Chi-squared
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Hydroxychloroquine; Test type: Superiority; p = 0.6617, Chi-squared
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Hydroxychloroquine; Test type: Superiority; p = 0.7309, Chi-squared
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Hydroxychloroquine; Test type: Superiority; p = 0.9861, Chi-squared

46. Primary Outcome: Number of Participants Who Met Medication Effectiveness Criteria: Adherence to Index Medication (Tofacitinib)
Description: Medication effectiveness criteria categorized as: 1) adherence to index medication, 2) no dose escalation for index medication, 3) no switch from index medication, 4) no addition of NB-DMARD, 5) criteria for oral glucocorticoids, 6) use of Injectable glucocorticoids. Adherence to index medication was defined as at least 30 days continuous supply of tofacitinib during post-index period.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 212 | 50 | 14
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.0880, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0065, Chi-squared

47. Primary Outcome: Number of Participants Who Met Medication Effectiveness Criteria: No Dose Escalation for Index Medication (Tofacitinib)
Description: Medication effectiveness criteria categorized as: 1) adherence to index medication, 2) no dose escalation for index medication, 3) no switch from index medication, 4) no addition of NB-DMARD, 5) criteria for oral glucocorticoids, 6) use of Injectable glucocorticoids. No dose escalation for index medication was defined as no increase in dose for index medication compared to the starting dose during post-index period.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 321 | 91 | 48
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.5157, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1231, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2109, Chi-squared

48. Primary Outcome: Number of Participants Who Met Medication Effectiveness Criteria: No Switch From Index Medication (Tofacitinib)
Description: Medication effectiveness criteria categorized as: 1) adherence to index medication, 2) no dose escalation for index medication, 3) no switch from index medication, 4) no addition of NB-DMARD, 5) criteria for oral glucocorticoids, 6) use of Injectable glucocorticoids. No switch from index medication was defined as no switching from the index medication to a (different) biologic agent during post-index period.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 273 | 77 | 36
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8424, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3278, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3336, Chi-squared

49. Primary Outcome: Number of Participants Who Met Medication Effectiveness Criteria: No Addition of NB-DMARD
Description: Medication effectiveness criteria categorized as: 1) adherence to index medication, 2) no dose escalation for index medication, 3) no switch from index medication, 4) no addition of NB-DMARD, 5) criteria for oral glucocorticoids, 6) use of Injectable glucocorticoids. No addition of NB-DMARD was defined as no addition of new NB-DMARD to index therapy during post-index period.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 319 | 84 | 46
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.0654, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7315, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1897, Chi-squared

50. Primary Outcome: Number of Participants Who Met Medication Effectiveness Criteria: Criteria for Oral Glucocorticoids
Description: Medication effectiveness criteria categorized as: 1) adherence to index medication, 2) no dose escalation for index medication, 3) no switch from index medication, 4) no addition of NB-DMARD, 5) criteria for oral glucocorticoids, 6) use of Injectable glucocorticoids. Medication effectiveness criteria for oral glucocorticoids was defined as either of the following: 1) Participants cannot receive oral glucocorticoids for > 30 days between (index date +91 days) to (index date + 359 days); 2) No increase in oral glucocorticoid dose during months 6-12 after index date.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 281 | 81 | 39
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.5146, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7121, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4434, Chi-squared

51. Primary Outcome: Number of Participants Who Met Medication Effectiveness Criteria: Use of Injectable Glucocorticoids
Description: Medication effectiveness criteria categorized as: 1) adherence to index medication, 2) no dose escalation for index medication, 3) no switch from index medication, 4) no addition of NB-DMARD, 5) criteria for oral glucocorticoids, 6) use of Injectable glucocorticoids. Use of Injectable glucocorticoids was defined as maximum one parenteral or intra-articular glucocorticoid joint injection use after the participant had been on biologic treatment for >3 months post index date ([index date +91 days] to [index date +359 days]).
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 278 | 77 | 36
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8966, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2105, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3336, Chi-squared

52. Primary Outcome: Number of Participants With All Cause Ambulatory Visits During Pre-Index Period
Description: Number of participants with at least one ambulatory visit that was due to all cause during the pre-index period is reported. All cause refers to ambulatory visits due to all comorbidities, including RA.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 337 | 94 | 48

53. Primary Outcome: Number of Participants With All Cause Emergency Department Visits During Pre-Index Period
Description: Number of participants with at least one emergency department visits that was due to all cause during the pre-index period is reported. All cause refers to emergency visits due to all comorbidities, including RA.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 88 | 29 | 15
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.3610, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4519, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.9612, Chi-squared

54. Primary Outcome: Number of Participants With All Cause Inpatient Admissions During Pre-Index Period
Description: Number of participants with at least one inpatient admissions that was due to all cause during the pre-index period is reported. All cause refers to inpatient admission due to all comorbidities, including RA.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 40 | 12 | 7
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8135, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.5910, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7635, Chi-squared

55. Primary Outcome: Number of Participants With RA Related Ambulatory Visits During Pre-Index Period
Description: Number of participants with at least one ambulatory visit that was due to RA during the pre-index period is reported. RA related refers to ambulatory visits due to RA.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 336 | 94 | 48
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.5970, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7055, Chi-squared

56. Primary Outcome: Number of Participants With RA Related Emergency Department Visits During Pre-Index Period
Description: Number of participants with at least one emergency department visits that was due to RA during the pre-index period is reported. RA related refers to emergency department visits due to RA.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 29 | 10 | 5
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.5435, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.6790, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.9676, Chi-squared

57. Primary Outcome: Number of Participants With RA Related Inpatient Admissions During Pre-Index Period
Description: Number of participants with at least one inpatient admissions that was due to RA during the pre-index period is reported. RA related refers to inpatient admission due to RA.
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 24 | 6 | 5
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8035, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.4184, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3950, Chi-squared

58. Primary Outcome: Number of Participants With All Cause Ambulatory Visits During Post-Index Period
Description: Number of participants with at least one ambulatory visit that was due to all cause during the post-index period is reported. All cause refers to ambulatory visits due to all comorbidities, including RA.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 337 | 94 | 48

59. Primary Outcome: Number of Participants With All Cause Emergency Department Visits During Post-Index Period
Description: Number of participants with at least one emergency department visits that was due to all cause during the post-index period is reported. All cause refers to emergency department visits due to all comorbidities, including RA.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 85 | 25 | 18
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.7871, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0722, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.1810, Chi-squared

60. Primary Outcome: Number of Participants With All Cause Inpatient Admissions During Post-Index Period
Description: Number of participants with at least one inpatient admissions that was due to all cause during the post-index period is reported. All cause refers to inpatient admissions due to all comorbidities, including RA.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 41 | 7 | 9
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.1984, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2043, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0439, Chi-squared

61. Primary Outcome: Number of Participants With RA Related Ambulatory Visits During Post Index Period
Description: Number of participants with at least one of the RA-related ambulatory visits during the post-index period is reported. RA related refers to ambulatory visits due to RA.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 335 | 92 | 48
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.1702, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.5926, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3088, Chi-squared

62. Primary Outcome: Number of Participants With RA Related Emergency Department Visits During Post Index Period
Description: Number of participants with at least one of the RA-related emergency department visit during the post-index period is reported. RA related refers to emergency department visits due to RA.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 24 | 7 | 4
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.9141, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7623, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.8517, Chi-squared

63. Primary Outcome: Number of Participants With RA Related Inpatient Admissions During Post Index Period
Description: Number of participants with at least one of an RA-related inpatient admission during the post-index period is reported. RA related refers to inpatient admissions due to RA.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
Participants | 31 | 4 | 9
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.1208, Chi-squared
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0425, Chi-squared
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0046, Chi-squared

64. Primary Outcome: Mean Total Health Care Cost All Cause During Pre-Index Period
Description: Mean total health care cost all cause during pre-index period is reported. All cause refers to cost spent due to all comorbidities including RA and calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs).
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars | 38294.06 (29855.01) | 37703.67 (34291.57) | 40845.52 (51582.10)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.8698, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7391, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.7043, t-test

65. Primary Outcome: Mean Total Health Care Cost RA Related During Pre-Index Period
Description: RA related healthcare cost refers to cost spent due to RA alone and was calculated as the total of treatment cost (cost of tofacitinib, biologic DMARDs, NB-DMARDs and administration of intravenous (IV) biologics) and medical cost (cost of ambulatory cost, emergency department visits cost, inpatient admission cost, home health care cost, urgent care cost and other medical services cost).
Time Frame: as for outcome 1
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars | 26310.56 (23044.42) | 21927.28 (18179.77) | 25941.25 (28226.04)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.0536, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.9313, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.3740, t-test

66. Primary Outcome: Mean Total Health Care Cost Due to All Cause During Post-Index Period
Description: Mean total health care cost due to all cause during post-index period is reported. All cause refers to cost spent due to all comorbidities, including RA and calculated as the total of pharmacy cost (cost of home healthcare cost, urgent care cost and other medical services costs) and medical cost (cost of ambulatory cost, emergency department visits cost, inpatient admission cost and other costs).
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars | 54792.79 (29936.57) | 52877.64 (44741.22) | 54617.88 (51150.03)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.6963, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.9816, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.8349, t-test

67. Primary Outcome: Mean Total Health Care Cost RA Related During Post-Index Period
Description: RA related healthcare cost refers to cost spent due to RA alone and was calculated as the total of treatment cost (cost of tofacitinib, biologic DMARDs, NB-DMARDs and administration of IV biologics) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost, home health care cost, urgent care cost and other medical services cost).
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars | 42402.93 (20786.01) | 35768.64 (13706.47) | 41984.33 (39638.80)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.0003, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.9431, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.2964, t-test

68. Primary Outcome: Mean Treatment Persistence Duration Measured for Index Medication (Tofacitinib)
Description: Treatment persistence with tofacitinib was defined as not having a gap in therapy of at least 60 days between prescription re-fills of tofacitinib.
Time Frame: as for outcome 13
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
days | 297.61 (99.42) | 284.48 (102.42) | 246.94 (120.12)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; Test type: Superiority; p = 0.2614, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0014, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; Test type: Superiority; p = 0.0535, t-test

69. Secondary Outcome: Mean Total All Cause Monthly Health Care Cost
Description: Mean total monthly health care cost due to all cause is reported. All cause refers to cost spent due to all comorbidities, including RA and calculated as the total of pharmacy cost (cost of home healthcare cost, urgent care cost and other medical services costs) and medical cost (cost of ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). Total all cause monthly health care cost is reported for every month from 12 months duration before index date (pre-index period) to 12 months duration post index date (post index period). Index date is defined as the date of first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During pre-index period (at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 months before index date) and post index period (at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 month post index date)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars
  1 month before index date | 1982.85 (3160.93) | 1298.00 (1660.83) | 1590.23 (2342.22)
  2 months before index date | 2961.52 (6134.21) | 2859.41 (4782.43) | 2007.33 (2279.76)
  3 months before index date | 2920.21 (3787.33) | 3160.66 (5286.29) | 2283.86 (2405.21)
  4 months before index date | 3218.67 (4385.35) | 3481.17 (4512.71) | 3255.21 (3927.64)
  5 months before index date | 3085.10 (4078.22) | 2821.69 (3482.77) | 4322.60 (12892.15)
  6 months before index date | 3708.45 (6412.35) | 3469.21 (7966.20) | 6210.48 (15934.47)
  7 months before index date | 3004.67 (3751.57) | 5219.03 (20901.31) | 3332.57 (4279.40)
  8 months before index date | 3650.97 (7165.39) | 3407.89 (6513.74) | 4578.01 (16218.40)
  9 months before index date | 3902.43 (7411.23) | 2798.05 (3916.34) | 4698.18 (13942.52)
  10 months before index date | 3128.19 (4655.37) | 3074.57 (5981.65) | 2850.71 (3512.63)
  11 months before index date | 3226.98 (6905.09) | 2765.39 (3795.95) | 2268.61 (2941.55)
  12 months before index date | 3504.01 (7280.54) | 3348.60 (7074.21) | 3447.74 (7167.30)
  1 month after index date | 6493.14 (5621.42) | 6219.90 (4771.10) | 5613.83 (2685.11)
  2 months after index date | 3401.05 (3629.35) | 3335.68 (2638.48) | 3534.10 (3435.08)
  3 months after index date | 5192.25 (12424.70) | 4274.36 (3929.19) | 7069.72 (23449.05)
  4 months after index date | 5542.45 (12928.65) | 3884.67 (2886.54) | 3936.05 (5042.01)
  5 months after index date | 3502.04 (5264.36) | 3164.43 (3257.78) | 3558.20 (4942.20)
  6 months after index date | 4367.35 (5250.44) | 3430.03 (4363.37) | 4062.60 (4741.14)
  7 months after index date | 4335.90 (5099.96) | 4876.01 (5517.19) | 6839.45 (24302.54)
  8 months after index date | 3998.48 (5427.41) | 3232.79 (3365.36) | 3870.33 (5967.14)
  9 months after index date | 4562.22 (7188.96) | 4250.44 (5153.79) | 3033.80 (4573.15)
  10 months after index date | 4680.99 (6427.93) | 4507.04 (4474.32) | 4208.68 (6898.73)
  11 months after index date | 4297.17 (5507.21) | 3527.33 (5467.69) | 3958.85 (6181.37)
  12 months after index date | 4419.74 (6361.66) | 8174.95 (40068.17) | 4932.28 (13927.49)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 1 months before index date; Test type: Superiority; p = 0.0051, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 months before index date; Test type: Superiority; p = 0.3041, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 months before index date; Test type: Superiority; p = 0.4432, t-test
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 2 months before index date; Test type: Superiority; p = 0.8641, t-test
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 months before index date; Test type: Superiority; p = 0.0435, t-test
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 months before index date; Test type: Superiority; p = 0.1530, t-test
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 months before index date; Test type: Superiority; p = 0.1188, t-test
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 3 months before index date; Test type: Superiority; p = 0.6807, t-test
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 months before index date; Test type: Superiority; p = 0.1772, t-test
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 4 months before index date; Test type: Superiority; p = 0.6104, t-test
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 months before index date; Test type: Superiority; p = 0.9564, t-test
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 months before index date; Test type: Superiority; p = 0.7688, t-test
Statistical Analysis 13: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 5 months before index date; Test type: Superiority; p = 0.5685, t-test
Statistical Analysis 14: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 months before index date; Test type: Superiority; p = 0.5122, t-test
Statistical Analysis 15: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 months before index date; Test type: Superiority; p = 0.4321, t-test
Statistical Analysis 16: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 6 months before index date; Test type: Superiority; p = 0.7892, t-test
Statistical Analysis 17: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 months before index date; Test type: Superiority; p = 0.2874, t-test
Statistical Analysis 18: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 months before index date; Test type: Superiority; p = 0.2662, t-test
Statistical Analysis 19: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 7 months before index date; Test type: Superiority; p = 0.3091, t-test
Statistical Analysis 20: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 months before index date; Test type: Superiority; p = 0.5783, t-test
Statistical Analysis 21: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 months before index date; Test type: Superiority; p = 0.4021, t-test
Statistical Analysis 22: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 8 months before index date; Test type: Superiority; p = 0.7670, t-test
Statistical Analysis 23: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 months before index date; Test type: Superiority; p = 0.6978, t-test
Statistical Analysis 24: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 months before index date; Test type: Superiority; p = 0.6328, t-test
Statistical Analysis 25: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 9 months before index date; Test type: Superiority; p = 0.0541, t-test
Statistical Analysis 26: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 months before index date; Test type: Superiority; p = 0.6999, t-test
Statistical Analysis 27: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 months before index date; Test type: Superiority; p = 0.3590, t-test
Statistical Analysis 28: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 10 months before index date; Test type: Superiority; p = 0.9360, t-test
Statistical Analysis 29: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 months before index date; Test type: Superiority; p = 0.6260, t-test
Statistical Analysis 30: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 months before index date; Test type: Superiority; p = 0.7797, t-test
Statistical Analysis 31: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 months before index date; Test type: Superiority; p = 0.0934, t-test
Statistical Analysis 32: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 11 months before index date; Test type: Superiority; p = 0.3960, t-test
Statistical Analysis 33: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 months before index date; Test type: Superiority; p = 0.4292, t-test
Statistical Analysis 34: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 12 months before index date; Test type: Superiority; p = 0.8540, t-test
Statistical Analysis 35: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 months before index date; Test type: Superiority; p = 0.9600, t-test
Statistical Analysis 36: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 months before index date; Test type: Superiority; p = 0.9374, t-test
Statistical Analysis 37: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 1 month after index date; Test type: Superiority; p = 0.6674, t-test
Statistical Analysis 38: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 month after index date; Test type: Superiority; p = 0.0776, t-test
Statistical Analysis 39: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 month after index date; Test type: Superiority; p = 0.3350, t-test
Statistical Analysis 40: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 2 month after index date; Test type: Superiority; p = 0.8461, t-test
Statistical Analysis 41: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 month after index date; Test type: Superiority; p = 0.8111, t-test
Statistical Analysis 42: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 month after index date; Test type: Superiority; p = 0.7267, t-test
Statistical Analysis 43: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 3 month after index date; Test type: Superiority; p = 0.2453, t-test
Statistical Analysis 44: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 month after index date; Test type: Superiority; p = 0.5889, t-test
Statistical Analysis 45: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 month after index date; Test type: Superiority; p = 0.4162, t-test
Statistical Analysis 46: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 4 month after index date; Test type: Superiority; p = 0.0307, t-test
Statistical Analysis 47: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 month after index date; Test type: Superiority; p = 0.1147, t-test
Statistical Analysis 48: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 month after index date; Test type: Superiority; p = 0.9481, t-test
Statistical Analysis 49: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 5 month after index date; Test type: Superiority; p = 0.4455, t-test
Statistical Analysis 50: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 month after index date; Test type: Superiority; p = 0.9445, t-test
Statistical Analysis 51: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 month after index date; Test type: Superiority; p = 0.6191, t-test
Statistical Analysis 52: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 6 month after index date; Test type: Superiority; p = 0.0805, t-test
Statistical Analysis 53: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 month after index date; Test type: Superiority; p = 0.7037, t-test
Statistical Analysis 54: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 month after index date; Test type: Superiority; p = 0.4288, t-test
Statistical Analysis 55: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 7 month after index date; Test type: Superiority; p = 0.3731, t-test
Statistical Analysis 56: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 month after index date; Test type: Superiority; p = 0.4803, t-test
Statistical Analysis 57: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 month after index date; Test type: Superiority; p = 0.5831, t-test
Statistical Analysis 58: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 8 month after index date; Test type: Superiority; p = 0.0944, t-test
Statistical Analysis 59: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 month after index date; Test type: Superiority; p = 0.8800, t-test
Statistical Analysis 60: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 month after index date; Test type: Superiority; p = 0.4949, t-test
Statistical Analysis 61: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 9 month after index date; Test type: Superiority; p = 0.6373, t-test
Statistical Analysis 62: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 month after index date; Test type: Superiority; p = 0.0497, t-test
Statistical Analysis 63: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 month after index date; Test type: Superiority; p = 0.1695, t-test
Statistical Analysis 64: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 month after index date; Test type: Superiority; p = 0.6373, t-test
Statistical Analysis 65: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 month after index date; Test type: Superiority; p = 0.7866, t-test
Statistical Analysis 66: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 10 months after index date; Test type: Superiority; p = 0.7643, t-test
Statistical Analysis 67: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 11 month after index date; Test type: Superiority; p = 0.2307, t-test
Statistical Analysis 68: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 month after index date; Test type: Superiority; p = 0.6712, t-test
Statistical Analysis 69: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 months after index date; Test type: Superiority; p = 0.6953, t-test
Statistical Analysis 70: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 12 month after index date; Test type: Superiority; p = 0.3675, t-test
Statistical Analysis 71: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 month after index date; Test type: Superiority; p = 0.8027, t-test
Statistical Analysis 72: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 month after index date; Test type: Superiority; p = 0.4817, t-test

70. Secondary Outcome: Mean Total RA Related Monthly Health Care Cost
Description: Mean total monthly health care cost due to RA is reported. RA related refers to cost spent by participants due to RA on health care services. This is calculated as the total of treatment cost (cost of tofacitinib, biologic DMARDs, NB-DMARDs and administration of IV biologics) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost, home health care cost, urgent care cost and other medical services cost). RA related monthly health care cost is reported for every month from 12 months duration before index date (pre-index period) to 12 months duration post index date (post index period). Index date is defined as the date of first claim for tofacitinib made by participants to their insurance provider during identification period of 3 years.
Time Frame: During pre-index period (at1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 months before index date) and post index period (at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 month after index date)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
Number analyzed (Participants) | 337 | 94 | 48
dollars
  1 month before index date | 1195.04 (2637.68) | 671.18 (1213.40) | 636.05 (1238.09)
  2 months before index date | 1903.16 (3155.45) | 1577.52 (2390.24) | 1141.74 (1700.28)
  3 months before index date | 2152.29 (3413.71) | 2361.03 (4927.73) | 1581.22 (2378.86)
  4 months before index date | 2168.50 (3489.71) | 2614.99 (4041.35) | 2285.37 (3322.71)
  5 months before index date | 2254.93 (3480.55) | 1917.28 (2766.38) | 3312.04 (12509.62)
  6 months before index date | 2422.23 (4000.01) | 1931.47 (3046.55) | 4535.86 (13927.05)
  7 months before index date | 2183.57 (3240.88) | 2403.88 (3808.44) | 1776.81 (2692.28)
  8 months before index date | 2697.28 (6295.30) | 1756.79 (2719.69) | 3511.39 (15412.06)
  9 months before index date | 2516.49 (4380.11) | 1700.46 (2463.15) | 1755.33 (2741.92)
  10 months before index date | 2420.82 (4487.55) | 1640.42 (2578.03) | 2197.70 (3256.25)
  11 months before index date | 1932.94 (3480.59) | 1664.42 (3182.62) | 1534.64 (2442.49)
  12 months before index date | 2463.30 (6488.79) | 1687.84 (2743.46) | 1673.11 (2538.14)
  1 month after index date | 5520.12 (3236.09) | 4864.96 (2427.19) | 5078.09 (2374.78)
  2 months after index date | 2475.97 (2565.47) | 2562.85 (1762.39) | 2467.49 (1841.74)
  3 months after index date | 4264.21 (11021.43) | 3525.69 (3579.91) | 5901.33 (22733.73)
  4 months after index date | 4513.18 (11997.33) | 3312.81 (2744.19) | 2193.74 (1997.44)
  5 months after index date | 2525.72 (3219.78) | 2171.23 (2225.60) | 2550.85 (4254.36)
  6 months after index date | 3448.44 (4479.50) | 2290.80 (2770.10) | 2715.92 (2695.20)
  7 months after index date | 3214.12 (3146.04) | 3172.63 (3093.67) | 6205.73 (23782.75)
  8 months after index date | 2792.29 (3675.52) | 2441.75 (2695.77) | 2888.44 (5532.83)
  9 months after index date | 3596.05 (6104.08) | 2667.32 (3922.25) | 2532.87 (4559.72)
  10 months after index date | 3536.10 (4403.21) | 3295.99 (3718.43) | 2521.96 (3201.05)
  11 months after index date | 3292.62 (4725.06) | 2574.32 (4803.21) | 2966.58 (5539.05)
  12 months after index date | 3224.11 (5151.51) | 2888.29 (4727.03) | 3961.34 (13543.17)
Statistical Analysis 1: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 1 month before index date; Test type: Superiority; p = 0.0063, t-test
Statistical Analysis 2: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 month before index date; Test type: Superiority; p = 0.0162, t-test
Statistical Analysis 3: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 month before index date; Test type: Superiority; p = 0.8715, t-test
Statistical Analysis 4: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 2 months before index date; Test type: Superiority; p = 0.2799, t-test
Statistical Analysis 5: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 months before index date; Test type: Superiority; p = 0.0126, t-test
Statistical Analysis 6: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 months before index date; Test type: Superiority; p = 0.2126, t-test
Statistical Analysis 7: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 3 months before index date; Test type: Superiority; p = 0.7004, t-test
Statistical Analysis 8: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 months before index date; Test type: Superiority; p = 0.1476, t-test
Statistical Analysis 9: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 months before index date; Test type: Superiority; p = 0.2057, t-test
Statistical Analysis 10: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 4 months before index date; Test type: Superiority; p = 0.2905, t-test
Statistical Analysis 11: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 months before index date; Test type: Superiority; p = 0.8273, t-test
Statistical Analysis 12: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 months before index date; Test type: Superiority; p = 0.6270, t-test
Statistical Analysis 13: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 5 months before index date; Test type: Superiority; p = 0.3256, t-test
Statistical Analysis 14: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 months before index date; Test type: Superiority; p = 0.5631, t-test
Statistical Analysis 15: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 months before index date; Test type: Superiority; p = 0.4491, t-test
Statistical Analysis 16: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 6 months before index date; Test type: Superiority; p = 0.2009, t-test
Statistical Analysis 17: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 months before index date; Test type: Superiority; p = 0.3011, t-test
Statistical Analysis 18: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 months before index date; Test type: Superiority; p = 0.2065, t-test
Statistical Analysis 19: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 7 months before index date; Test type: Superiority; p = 0.6098, t-test
Statistical Analysis 20: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 months before index date; Test type: Superiority; p = 0.2586, t-test
Statistical Analysis 21: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 months before index date; Test type: Superiority; p = 0.4074, t-test
Statistical Analysis 22: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 8 months before index date; Test type: Superiority; p = 0.0345, t-test
Statistical Analysis 23: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 months before index date; Test type: Superiority; p = 0.4377, t-test
Statistical Analysis 24: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 months before index date; Test type: Superiority; p = 0.7191, t-test
Statistical Analysis 25: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 9 months before index date; Test type: Superiority; p = 0.0199, t-test
Statistical Analysis 26: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 months before index date; Test type: Superiority; p = 0.1032, t-test
Statistical Analysis 27: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 months before index date; Test type: Superiority; p = 0.9040, t-test
Statistical Analysis 28: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 10 months before index date; Test type: Superiority; p = 0.0316, t-test
Statistical Analysis 29: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 months before index date; Test type: Superiority; p = 0.6748, t-test
Statistical Analysis 30: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 months before index date; Test type: Superiority; p = 0.2679, t-test
Statistical Analysis 31: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 11 months before index date; Test type: Superiority; p = 0.5010, t-test
Statistical Analysis 32: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 months before index date; Test type: Superiority; p = 0.3228, t-test
Statistical Analysis 33: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 months before index date; Test type: Superiority; p = 0.7881, t-test
Statistical Analysis 34: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 12 months before index date; Test type: Superiority; p = 0.0876, t-test
Statistical Analysis 35: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 months before index date; Test type: Superiority; p = 0.1226, t-test
Statistical Analysis 36: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 months before index date; Test type: Superiority; p = 0.9753, t-test
Statistical Analysis 37: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 1 month after index date; Test type: Superiority; p = 0.0336, t-test
Statistical Analysis 38: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 month after index date; Test type: Superiority; p = 0.2551, t-test
Statistical Analysis 39: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 1 month after index date; Test type: Superiority; p = 0.6189, t-test
Statistical Analysis 40: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 2 months after index date; Test type: Superiority; p = 0.7051, t-test
Statistical Analysis 41: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 months after index date; Test type: Superiority; p = 0.9775, t-test
Statistical Analysis 42: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 2 months after index date; Test type: Superiority; p = 0.7643, t-test
Statistical Analysis 43: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 3 months after index date; Test type: Superiority; p = 0.2953, t-test
Statistical Analysis 44: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 months after index date; Test type: Superiority; p = 0.6257, t-test
Statistical Analysis 45: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 3 months after index date; Test type: Superiority; p = 0.4753, t-test
Statistical Analysis 46: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 4 months after index date; Test type: Superiority; p = 0.0926, t-test
Statistical Analysis 47: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 months after index date; Test type: Superiority; p = 0.0013, t-test
Statistical Analysis 48: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 4 months after index date; Test type: Superiority; p = 0.0065, t-test
Statistical Analysis 49: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 5 months after index date; Test type: Superiority; p = 0.2212, t-test
Statistical Analysis 50: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 months after index date; Test type: Superiority; p = 0.9688, t-test
Statistical Analysis 51: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 5 months after index date; Test type: Superiority; p = 0.5647, t-test
Statistical Analysis 52: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 6 months after index date; Test type: Superiority; p = 0.0023, t-test
Statistical Analysis 53: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 months after index date; Test type: Superiority; p = 0.1142, t-test
Statistical Analysis 54: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 6 months after index date; Test type: Superiority; p = 0.3842, t-test
Statistical Analysis 55: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 7 months after index date; Test type: Superiority; p = 0.9097, t-test
Statistical Analysis 56: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 months after index date; Test type: Superiority; p = 0.3885, t-test
Statistical Analysis 57: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 7 months after index date; Test type: Superiority; p = 0.3834, t-test
Statistical Analysis 58: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 8 months after index date; Test type: Superiority; p = 0.3075, t-test
Statistical Analysis 59: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 months after index date; Test type: Superiority; p = 0.9075, t-test
Statistical Analysis 60: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 8 months after index date; Test type: Superiority; p = 0.5993, t-test
Statistical Analysis 61: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 9 months after index date; Test type: Superiority; p = 0.0775, t-test
Statistical Analysis 62: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 months after index date; Test type: Superiority; p = 0.1536, t-test
Statistical Analysis 63: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 9 months after index date; Test type: Superiority; p = 0.8553, t-test
Statistical Analysis 64: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 10 months after index date; Test type: Superiority; p = 0.6295, t-test
Statistical Analysis 65: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 months after index date; Test type: Superiority; p = 0.0551, t-test
Statistical Analysis 66: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 10 months after index date; Test type: Superiority; p = 0.2215, t-test
Statistical Analysis 67: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 11 months after index date; Test type: Superiority; p = 0.1948, t-test
Statistical Analysis 68: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 months after index date; Test type: Superiority; p = 0.6621, t-test
Statistical Analysis 69: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 11 months after index date; Test type: Superiority; p = 0.6629, t-test
Statistical Analysis 70: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Discontinued; 12 months after index date; Test type: Superiority; p = 0.5699, t-test
Statistical Analysis 71: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Persistent vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 months after index date; Test type: Superiority; p = 0.7105, t-test
Statistical Analysis 72: Comparison: Methotrexate (MTX) + Tofacitinib: MTX Discontinued vs Methotrexate (MTX) + Tofacitinib: MTX Interrupted; 12 months after index date; Test type: Superiority; p = 0.5965, t-test

ADVERSE EVENTS:
Description: Due to the nature of claims data base from which these data where queried, no adverse events were collected in this study.
Arm/Group | Methotrexate (MTX) + Tofacitinib: MTX Persistent | Methotrexate (MTX) + Tofacitinib: MTX Discontinued | Methotrexate (MTX) + Tofacitinib: MTX Interrupted
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03975790/Prot_SAP_000.pdf